CLINICAL TRIAL: NCT00937326
Title: A Phase II, Randomized, Placebo-Controlled, Double-Blind, Multiple-Dose Clinical Study to Assess the Safety and Pharmacokinetics of SRT2104 in Type 2 Diabetic Human Subjects
Brief Title: Clinical Study to Assess the Safety and Pharmacokinetics of SRT2104 in Type 2 Diabetic Human Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sirtris, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 113160
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SRT2104

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): The Placebo treatment group will be administered eight placebo capsules per day.
  Placebo will be administered orally once daily for twenty-eight consecutive days. Dosing will take place at approximately the same time every morning, approximately 15 minutes following consumption of a standardized meal and should be administered with approximately 1 to 2 glasses of water.
  Interventions: Drug: Placebo
- Arm1 - 0.25g (Active Comparator): The 0.25g SRT2104 treatment group will be administered one SRT2104 capsules with 7 placebo capsules, for a total of 8 capsules per day.
  0.25g SRT2104 will be administered orally once daily for twenty-eight consecutive days. Dosing will take place at approximately the same time every morning, 15 minutes following consumption of a standardized meal and should be administered with approximately 1 to 2 glasses of water.
  Interventions: Drug: SRT2104; Drug: Placebo
- Arm2 - 0.5g (Active Comparator): The 0.5g SRT2104 treatment group will be administered two SRT2104 capsules with 6 placebo capsules, for a total of 8 capsules per day.
  0.5g SRT2104 will be administered orally once daily for twenty-eight consecutive days. Dosing will take place at approximately the same time every morning, 15 minutes following consumption of a standardized meal and should be administered with approximately 1 to 2 glasses of water.
  Interventions: Drug: SRT2104; Drug: Placebo
- Arm3 - 1g (Active Comparator): The 1g SRT2104 treatment group will be administered four SRT2104 capsules with four placebo capsules, for a total of 8 capsules per day.
  1g SRT2104 will be administered orally once daily for twenty-eight consecutive days. Dosing will take place at approximately the same time every morning, 15 minutes following consumption of a standardized meal and should be administered with approximately 1 to 2 glasses of water.
  Interventions: Drug: SRT2104; Drug: Placebo
- Arm4 - 2g (Active Comparator): The 2g SRT2104 treatment group will be administered eight SRT2104 capsules per day.
  2g SRT2104 will be administered orally once daily for twenty-eight consecutive days. Dosing will take place at approximately the same time every morning, 15 minutes following consumption of a standardized meal and should be administered with approximately 1 to 2 glasses of water.
  Interventions: Drug: SRT2104

INTERVENTIONS:
Drug: SRT2104 — SRT2104 will be supplied as hard gelatin capsules, with each containing 250 mg.
  Arms: Arm1 - 0.25g; Arm2 - 0.5g; Arm3 - 1g; Arm4 - 2g
Drug: Placebo — Placebo will be supplied as hard gelatin capsules, with each containing an appropriate amount of placebo.
  Arms: Arm1 - 0.25g; Arm2 - 0.5g; Arm3 - 1g; Placebo

SUMMARY:
The primary purpose of this study is to determine the safety and tolerability of SRT2104 (0.25, 0.5, 1.0, and 2.0 g/day) in type 2 diabetic subjects when administered once daily for 28 consecutive days, and to characterize the pharmacokinetic profile of SRT2104 after a single dose and multiple administrations in type 2 diabetic subjects.

The secondary purpose of this study is to determine the effect of SRT2104 (0.25, 0.5, 1.0, and 2.0 g/day) when administered once daily for 28 consecutive days on fasting blood glucose and insulin and post-prandial blood glucose and insulin in type 2 diabetic subjects.

DETAILED DESCRIPTION:
Study Objectives

Primary:

1. To determine the safety and tolerability of SRT2104 (0.25, 0.5, 1.0, and 2.0 g/day) in type 2 diabetic subjects when administered once daily for 28 consecutive days.
2. To characterize the pharmacokinetic profile of SRT2104 (0.25, 0.5, 1.0, and 2.0 g/day) after a single dose and multiple administrations in type 2 diabetic subjects.

Secondary:

1. To determine the effect of SRT2104 (0.25, 0.5, 1.0, and 2.0 g/day) when administered once daily for 28 consecutive days on fasting blood glucose and insulin and post-prandial blood glucose and insulin in type 2 diabetic subjects.

Study Design:

Prospective, multi-center, clinical study of SRT2104 administered orally once daily for 28 consecutive days; randomized, placebo-controlled, double-blind, multiple-dose, inpatient/outpatient study to assess the safety and pharmacokinetics (PK) of SRT2104 in type 2 diabetic male and female subjects on an existing, stable, background metformin therapy. Approximately 225 subjects aged 30-70, who fulfill the inclusion/exclusion criteria, will be enrolled in this study to ensure completion of forty (40) evaluable subjects within each of five dosing groups. Subjects will be evenly randomized to receive SRT2104 at one of five doses, placebo (A), 0.25 g/day (B), 0.5 g/day (C), 1.0 g/day (D), or 2.0 g/day (E), once a day for 28 consecutive days, approximately 15 minutes following consumption of a standardized meal. Subjects will remain on a fixed dose of test material for all dosing days in the study.

Subjects will sign the informed consent form at the Screening Visit, and will undergo screening assessments over a 2-day period to verify eligibility for the study. If eligible and willing to participate, subjects will return to the clinic within 21 days of the Screening Visit to participate in the dosing phase of the study. Subjects will be randomized to receive SRT2104 or placebo, and will be required to stay overnight at the study center on Day -1 and Day 27 to gather required PK samples and to assess safety on Day 1 and Day 28 respectively. In addition, subjects will be asked to return to the study center on Days 2 and 29; for three interim weekly safety assessments (on Days 8, 15, 22); and for an End of Study safety assessment 7 days after they complete the 28-day dosing period. A follow-up safety call will be made to each subject 30 days following their final dose of SRT2104 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of any race and gender within the age range of 30 to 70 years.
2. All female subjects must be of non-child-bearing potential. For the purposes of this study, this is defined as the subject being amenorrheic for at least 12 consecutive months, or at least 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy, or women who underwent tubal ligation. Menopausal status will be confirmed by demonstrating levels of follicle stimulating hormone (FSH) 40 - 138 mIU/ml and oestradiol < 20 pg/ml at entry, unless this information is available in the subject's medical record. In the event a subject's menopause status has been clearly established (for example, the subject indicates she has been amenorrheic for 10 years), but FSH and/or oestradiol levels are not consistent with a post-menopausal condition, determination of subject eligibility will be at the discretion of the principal investigator following consultation with the sponsor and medical monitor
3. All male subjects must agree with their partners to use double-barrier birth control or abstinence while participating in the study and for 12 weeks following the last dose of study drug.
4. Willingness to provide written informed consent to participate in the study
5. HbA1c ≥ 7.5 and ≤ 10.5
6. Fasting glucose ≥ 160 and ≤ 240 mg/dL
7. Body Mass Index (BMI) ≥ 25.0 kg/m^2 and ≤ 40.0 kg/m^2
8. On stable metformin medication for at least 3 months (≥ 1.0 g/day) prior to Screening
9. No prior history of HIV 1 or 2
10. Absence of disease markers for hepatitis B & C virus
11. Absence of significant disease or clinically significant abnormal laboratory values on the laboratory evaluations, medical history or physical examination during the screening; normal end organ function
12. Have a normal 12-lead ECG or one with abnormality considered to be clinically insignificant
13. Have a normal chest X-ray (P. A. View) or one with abnormality considered to be clinically insignificant
14. Comprehension of the nature and purpose of the study and compliance with the requirement of the entire protocol

Exclusion Criteria:

1. Any major illness in the past three months or any significant ongoing chronic medical illness not related to diabetes
2. Renal or liver impairment, defined as serum creatinine level of ≥ 1.4 mg/dL for females and ≥ 1.5 mg/dL for males, and greater than two times the upper limit of normal for liver enzymes, respectively.
3. History of or current gastro-intestinal diseases influencing drug absorption, except for appendectomy
4. History, within 3 years, of drug abuse (including Benzodiazepines, opioids, amphetamine, cocaine, and THC)
5. History of alcoholism (more than two years), moderate drinkers (more than three drinks per day) or having consumed alcohol within 48 hrs prior to dosing [one drink is equal to one unit of alcohol (one glass wine, half pint beer, one measure of spirit)]
6. Participation in any clinical trial within the past three months
7. History of difficulty in donating blood or accessibility of veins in left or right arm
8. Donation of blood (one unit or 350 ml) within three months prior to receiving the first dose of test material
9. Use of any prescription drug therapy, with exception of any prescription medication administered at a stable dose for at least 6 weeks prior to Screening, provided the medication is not contraindicated by the metformin label
10. Use of any alternate anti-diabetic therapy, except metformin, within three months of enrollment

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2009-08-19 (Actual); Primary Completion 2010-09-18 (Actual); Study Completion 2010-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (48):
- Bulgaria (7):
  - GSK Investigational Site, Byala
  - GSK Investigational Site, Dimitrovgrad
  - GSK Investigational Site, Haskovo
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
- GSK Investigational Site, Tallinn, Estonia
- Hungary (7):
  - GSK Investigational Site, Balantonfured
  - GSK Investigational Site, Eger
  - GSK Investigational Site, Gyula
  - GSK Investigational Site, Kecskemét
  - GSK Investigational Site, Sopron
  - GSK Investigational Site, Szekszárd
  - GSK Investigational Site, Zalaegerszeg
- Poland (8):
  - GSK Investigational Site, Cieszyn
  - GSK Investigational Site, Lubin
  - GSK Investigational Site, Puławy
  - GSK Investigational Site, Radzymin
  - GSK Investigational Site, Ruda Śląska
  - GSK Investigational Site, Słupsk
  - GSK Investigational Site, Tychy
  - GSK Investigational Site, Warsaw
- Romania (7):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Brăila
  - GSK Investigational Site, Buzău
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Oradea
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Timișoara
- Russia (9):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Rostov-on-Don
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tyumen
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Yaroslavl
- Ukraine (6):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Mykolaiv
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Ternopil
  - GSK Investigational Site, Vinnitsa
  - GSK Investigational Site, Zaporizhzhya
- United Kingdom (3):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, London
  - GSK Investigational Site, Newport

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 113160 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113160 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113160 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113160 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113160 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113160 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113160 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned on 225 male and female participants with type 2 diabetes (T2D) on an existing, stable, background metformin therapy, aged 30 to 70 years, at 45 centers of Bulgaria (7), Estonia (1), Hungary (4), Poland (4), Romania (6), Russia (13), United Kingdom (3) and Ukraine (7) from 19 August 2009 to 18 September 2010.
Pre-assignment Details: Out of 527 participants screened, 227 with glycosylated hemoglobin A (HbA1c) of >=7.5% and <= 10.5% and a fasting glucose (FG) >=160 and <=240 milligram per deciliter (mg/dL) were randomized in 1:1:1:1:1 to oral dose of placebo or any one of 4 doses of SRT2104 (0.25, 0.5, 1.0 or 2.0 gram per day [g/day]), once a day for 28 consecutive days.
Groups:
- Placebo: Participants received oral dose of matching placebo to SRT2104 capsule, once daily for 28 consecutive days. The study medication was administered as 8 capsules per day to maintain the blinding, at the same time every morning, approximately 15-30 minutes (min) following the start of meal consumption with 1 to 2 glasses of water.
- SRT2104 0.25 g/Day: Participants received oral dose of SRT2104 0.25 g/day capsule, once daily for 28 consecutive days. The study medication was administered as 8 capsules per day to maintain the blinding, at the same time every morning, approximately 15-30 min following the start of meal consumption with 1 to 2 glasses of water.
- SRT2104 0.5 g/Day: Participants received oral dose of SRT2104 0.5 g/day capsule, once daily for 28 consecutive days. The study medication was administered as 8 capsules per day to maintain the blinding, at the same time every morning, approximately 15-30 min following the start of meal consumption with 1 to 2 glasses of water.
- SRT2104 1.0 g/Day: Participants received oral dose of SRT2104 1.0 g/day capsule, once daily for 28 consecutive days. The study medication was administered as 8 capsules per day to maintain the blinding, at the same time every morning, approximately 15-30 min following the start of meal consumption with 1 to 2 glasses of water.
- SRT2104 2.0 g/Day: Participants received oral dose of SRT2104 2.0 g/day capsule, once daily for 28 consecutive days. The study medication was administered as 8 capsules per day to maintain the blinding, at the same time every morning, approximately 15-30 min following the start of meal consumption with 1 to 2 glasses of water.
Period: Overall Study
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Started | 46 | 45 | 46 | 45 | 45
Completed | 43 | 38 | 42 | 40 | 40
Not Completed | 3 | 7 | 4 | 5 | 5
Not completed — Adverse Event | 0 | 3 | 1 | 1 | 2
Not completed — Death | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 1 | 4 | 3
Not completed — Chest X-ray showed a suspicious shadow | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received oral dose of matching placebo to SRT2104 capsule, once daily for 28 consecutive days. The study medication was administered as 8 capsules per day to maintain the blinding, at the same time every morning, approximately 15-30 min following the start of meal consumption with 1 to 2 glasses of water.
- Total: Total of all reporting groups
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day | Total
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45 | 227
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.8 (8.40) | 58.2 (8.04) | 57.7 (9.00) | 57.3 (8.95) | 55.9 (9.03) | 57.0 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 22 | 28 | 30 | 18 | 126
  Male | 18 | 23 | 18 | 15 | 27 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1
  White | 45 | 45 | 46 | 45 | 44 | 225
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE), Serious Adverse Event (SAE), AE Related to Study Medication, AE Leading to Discontinuation and Fatal AE of Death
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition. AE's were classified as related to the study medication, based on the investigator's judgment.
Time Frame: Up to Follow-up (58 days)
Population: Safety Analysis Set (SAF) Population was defined as all participants who received at least one dose of any test material during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Participants
  Any AE | 11 | 15 | 19 | 11 | 15
  Any SAE | 0 | 1 | 1 | 0 | 0
  Any AE related to study medication | 0 | 1 | 0 | 1 | 1
  Any AE leading to discontinuation | 0 | 3 | 2 | 1 | 2
  Any fatal AE of death | 0 | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day in number of participants with any AE; Test type: Superiority; p = 0.4816, Fisher Exact — No adjustments for covariates were made
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day in number of participants with any AE; Test type: Superiority; p = 0.1147, Fisher Exact — No adjustments for covariates were made
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day in number of participants with any AE; Test type: Superiority; p = 1.0000, Fisher Exact — No adjustments for covariates were made
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day in number of participants with any AE; Test type: Superiority; p = 0.4816, Fisher Exact — No adjustments for covariates were made

2. Primary Outcome: Number of Participants With AE by Intensity of Mild, Moderate and Severe
Description: Intensity for each AE was categorized as mild, moderate and severe. Mild was defined as awareness of sign or symptom, but easily tolerated; moderate was defined as discomfort enough to cause interference with normal daily activities; severe was defined as inability to perform normal daily activities.
Time Frame: Up to Follow-up (58 days)
Population: Safety Analysis Set Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Participants
  Mild AE | 8 | 10 | 11 | 8 | 9
  Moderate AE | 7 | 6 | 12 | 5 | 7
  Severe AE | 0 | 1 | 1 | 0 | 0

3. Primary Outcome: Mean Change From Baseline in Weight Over Time
Description: Participant's body weight was assessed in the beginning of the study (at Day 1) and at the end of the study (Day 28 and Day 35). The clinical staff was instructed to use calibrated scales for weight measurement. The same scale was used at the clinical site for all participants at each specified time point during the study. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Kilogram (kg)
  Day 28: number analyzed (Participants) | 42 | 37 | 42 | 40 | 39
  Day 28 | -0.17 (1.25) | -0.81 (2.21) | -1.25 (2.06) | -0.56 (1.68) | -1.54 (3.82)
  Day 35: number analyzed (Participants) | 42 | 41 | 41 | 39 | 39
  Day 35 | -0.40 (1.39) | -0.91 (2.90) | -1.32 (1.89) | -0.86 (1.78) | -2.74 (7.27)

4. Primary Outcome: Change From Baseline in Vital Sign Parameter of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Over Time
Description: Vital sign assessment of SBP and DBP was done at Day 1 (pre-dose, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours and 24 hours post-dose), Day 2 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 8 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 15 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 22 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 27, Day 28 (pre-dose, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours and 24 hours post-dose) and Day 35. A window of plus or minus 5 minutes was allowed during the active treatment visit vital sign assessments. Baseline was defined as the assessment done on Day 1 (pre-dose). The change from Baseline was calculated by subtracting the Baseline value (Day 1, pre-dose) from the individual post-Baseline (Day 1, Day 2, Day 8, Day 15, Day 22, Day 27, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1, pre-dose) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Millimeter of mercury (mmHg)
  SBP, Day 1, 15 minutes: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  SBP, Day 1, 15 minutes | -1.49 (9.45) | 1.30 (8.36) | 0.36 (5.27) | -0.88 (5.13) | -0.24 (5.45)
  SBP, Day 1, 30 minutes: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  SBP, Day 1, 30 minutes | -1.44 (7.16) | 0.02 (6.24) | 1.36 (5.59) | -0.95 (6.05) | -1.10 (6.80)
  SBP, Day 1, 1 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  SBP, Day 1, 1 hour | -2.51 (10.03) | -0.81 (6.78) | -0.02 (6.33) | -1.83 (5.68) | -1.40 (7.11)
  SBP, Day 1, 2 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  SBP, Day 1, 2 hour | -1.60 (10.25) | -0.51 (5.51) | -1.45 (7.30) | -1.64 (7.51) | -2.93 (7.77)
  SBP, Day 1, 3 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  SBP, Day 1, 3 hour | -2.33 (10.78) | -1.14 (5.58) | -1.98 (7.22) | -1.33 (6.61) | -2.71 (7.61)
  SBP, Day 1, 4 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  SBP, Day 1, 4 hour | -3.51 (11.38) | -1.53 (6.52) | -0.86 (7.33) | -3.71 (8.71) | -2.74 (8.16)
  SBP, Day 1, 8 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  SBP, Day 1, 8 hour | -4.07 (9.19) | -0.93 (7.06) | 0.39 (6.96) | -2.26 (8.50) | -1.45 (7.23)
  SBP, Day 1, 12 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  SBP, Day 1, 12 hour | -3.02 (12.64) | 0.02 (7.63) | 0.02 (7.78) | -0.83 (8.30) | 0.81 (8.03)
  SBP, Day 1, 24 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  SBP, Day 1, 24 hour | -1.41 (6.11) | 0.14 (4.75) | -0.44 (5.68) | -0.02 (5.26) | -1.39 (6.21)
  SBP, Day 2, pre-dose: number analyzed (Participants) | 42 | 43 | 43 | 42 | 42
  SBP, Day 2, pre-dose | -1.64 (8.49) | -0.30 (6.49) | -1.05 (6.85) | -0.31 (6.79) | -2.50 (7.70)
  SBP, Day 2, 5 minutes: number analyzed (Participants) | 42 | 43 | 41 | 42 | 42
  SBP, Day 2, 5 minutes | -2.81 (9.74) | -0.47 (7.07) | -0.54 (5.78) | -0.40 (6.67) | -1.45 (8.00)
  SBP, Day 2, 30 minutes: number analyzed (Participants) | 38 | 40 | 38 | 41 | 40
  SBP, Day 2, 30 minutes | -3.13 (8.79) | -0.43 (6.81) | -1.47 (5.99) | -2.00 (6.88) | -1.38 (6.88)
  SBP, Day 2, 1 hour: number analyzed (Participants) | 37 | 40 | 38 | 41 | 40
  SBP, Day 2, 1 hour | -3.22 (8.67) | -0.48 (6.24) | -1.34 (7.33) | -1.32 (7.67) | -0.88 (7.38)
  SBP, Day 8, pre-dose: number analyzed (Participants) | 42 | 43 | 43 | 41 | 39
  SBP, Day 8, pre-dose | -2.83 (10.96) | -1.63 (6.22) | 0.42 (10.22) | 0.68 (9.93) | -1.36 (8.57)
  SBP, Day 8, 5 minutes: number analyzed (Participants) | 42 | 43 | 42 | 41 | 40
  SBP, Day 8, 5 minutes | -3.67 (10.94) | -1.47 (5.50) | 1.00 (7.76) | 1.20 (9.63) | -0.73 (7.93)
  SBP, Day 8, 30 minutes: number analyzed (Participants) | 39 | 40 | 38 | 40 | 38
  SBP, Day 8, 30 minutes | -1.72 (9.10) | -0.85 (6.48) | -0.29 (7.82) | 0.33 (9.31) | -1.92 (8.31)
  SBP, Day 8, 1 hour: number analyzed (Participants) | 38 | 40 | 38 | 40 | 38
  SBP, Day 8, 1 hour | -2.24 (10.22) | -1.00 (5.68) | -1.71 (7.80) | -2.75 (10.30) | -1.87 (7.66)
  SBP, Day 15, pre-dose: number analyzed (Participants) | 43 | 40 | 43 | 41 | 40
  SBP, Day 15, pre-dose | -2.77 (10.88) | -0.43 (7.22) | 0.65 (8.22) | 0.76 (9.66) | 0.03 (8.50)
  SBP, Day 15, 5 minutes: number analyzed (Participants) | 43 | 40 | 42 | 41 | 40
  SBP, Day 15, 5 minutes | -4.16 (12.17) | -1.15 (6.47) | 0.69 (8.67) | -0.27 (7.89) | -1.18 (8.75)
  SBP, Day 15, 30 minutes: number analyzed (Participants) | 39 | 38 | 39 | 41 | 38
  SBP, Day 15, 30 minutes | -3.56 (10.28) | -0.61 (8.31) | 0.03 (8.98) | -1.83 (9.16) | -1.97 (8.36)
  SBP, Day 15, 1 hour: number analyzed (Participants) | 38 | 37 | 39 | 41 | 38
  SBP, Day 15, 1 hour | -3.50 (10.25) | -0.24 (6.43) | -0.54 (7.27) | -0.98 (9.96) | -1.50 (7.91)
  SBP, Day 22, pre-dose: number analyzed (Participants) | 43 | 39 | 43 | 40 | 39
  SBP, Day 22, pre-dose | -2.07 (9.75) | -0.67 (8.49) | -0.53 (8.71) | -0.08 (9.92) | 0.08 (10.59)
  SBP, Day 22, 5 minutes: number analyzed (Participants) | 43 | 39 | 42 | 40 | 39
  SBP, Day 22, 5 minutes | -3.77 (11.97) | -1.46 (6.87) | -0.57 (6.72) | 0.08 (9.18) | -1.18 (9.91)
  SBP, Day 22, 30 minutes: number analyzed (Participants) | 39 | 36 | 39 | 40 | 37
  SBP, Day 22, 30 minutes | -3.03 (10.05) | -1.56 (6.64) | -1.77 (6.69) | -1.10 (9.78) | -2.05 (8.73)
  SBP, Day 22, 1 hour: number analyzed (Participants) | 38 | 36 | 39 | 40 | 37
  SBP, Day 22, 1 hour | -3.39 (9.31) | -1.64 (6.68) | -1.51 (8.29) | -0.85 (9.57) | -2.24 (9.37)
  SBP, Day 27: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  SBP, Day 27 | -2.91 (9.87) | -0.49 (7.74) | -0.48 (8.68) | 0.15 (9.04) | -1.05 (8.69)
  SBP, Day 28, pre-dose: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  SBP, Day 28, pre-dose | -2.60 (10.39) | -0.05 (7.17) | -1.10 (9.35) | 0.70 (9.92) | -0.90 (8.04)
  SBP, Day 28, 15 minutes: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  SBP, Day 28, 15 minutes | -4.58 (11.88) | -1.86 (7.11) | -1.21 (9.99) | -0.63 (9.60) | -1.56 (8.34)
  SBP, Day 28, 30 minutes: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  SBP, Day 28, 30 minutes | -4.07 (11.26) | -2.65 (6.47) | -1.69 (9.70) | -1.43 (9.09) | -2.44 (8.02)
  SBP, Day 28, 1 hour: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  SBP, Day 28, 1 hour | -4.74 (11.62) | -2.78 (6.77) | -1.26 (8.40) | -2.13 (9.24) | -3.85 (7.35)
  SBP, Day 28, 2 hour: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  SBP, Day 28, 2 hour | -5.07 (12.33) | -2.65 (6.63) | -0.98 (9.10) | -2.90 (7.32) | -3.21 (8.70)
  SBP, Day 28, 3 hour: number analyzed (Participants) | 42 | 37 | 42 | 40 | 39
  SBP, Day 28, 3 hour | -4.33 (11.33) | -2.84 (6.24) | -2.60 (8.32) | -2.03 (8.98) | -1.79 (9.01)
  SBP, Day 28, 4 hour: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  SBP, Day 28, 4 hour | -4.28 (11.36) | -3.16 (6.86) | -2.21 (7.89) | -3.48 (9.35) | -2.21 (7.56)
  SBP, Day 28, 8 hour: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  SBP, Day 28, 8 hour | -4.51 (12.32) | -2.11 (7.12) | -1.45 (8.96) | -2.83 (9.35) | -1.85 (9.02)
  SBP, Day 28, 12 hour: number analyzed (Participants) | 43 | 38 | 42 | 40 | 39
  SBP, Day 28, 12 hour | -4.95 (11.61) | -0.97 (6.73) | -2.14 (8.08) | -0.75 (8.48) | -0.82 (9.52)
  SBP, Day 28, 24 hour: number analyzed (Participants) | 43 | 38 | 42 | 40 | 39
  SBP, Day 28, 24 hour | -4.05 (11.72) | -1.42 (6.82) | -1.45 (7.42) | -0.08 (8.02) | -3.00 (8.28)
  SBP, Day 35: number analyzed (Participants) | 43 | 42 | 43 | 41 | 41
  SBP, Day 35 | -4.44 (12.39) | -2.83 (7.47) | -0.70 (8.05) | 0.37 (8.66) | -0.51 (9.88)
  DBP, Day 1, 15 minutes: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  DBP, Day 1, 15 minutes | -1.12 (6.71) | -0.42 (5.13) | -1.41 (6.44) | -0.38 (5.96) | -1.55 (5.67)
  DBP, Day 1, 30 minutes: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  DBP, Day 1, 30 minutes | -1.37 (5.98) | -1.05 (4.35) | -1.73 (5.87) | -0.29 (5.75) | -1.88 (5.87)
  DBP, Day 1, 1 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  DBP, Day 1, 1 hour | -2.70 (6.65) | -1.09 (5.12) | -1.89 (5.91) | -0.95 (5.64) | -2.83 (5.33)
  DBP, Day 1, 2 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  DBP, Day 1, 2 hour | -0.74 (7.50) | -1.26 (6.08) | -1.66 (5.69) | -0.45 (5.32) | -3.55 (6.01)
  DBP, Day 1, 3 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  DBP, Day 1, 3 hour | -1.74 (6.08) | -1.28 (6.03) | -2.57 (5.60) | -1.81 (6.73) | -1.76 (5.13)
  DBP, Day 1, 4 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  DBP, Day 1, 4 hour | -1.86 (7.88) | -0.77 (6.56) | -2.00 (6.46) | -0.90 (6.81) | -1.69 (5.05)
  DBP, Day 1, 8 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  DBP, Day 1, 8 hour | -2.16 (6.91) | -0.56 (6.42) | -0.73 (6.23) | -1.98 (6.23) | -1.52 (6.69)
  DBP, Day 1, 12 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  DBP, Day 1, 12 hour | -1.40 (8.76) | -0.16 (7.16) | -1.64 (7.81) | -1.24 (6.14) | -0.38 (5.78)
  DBP, Day 1, 24 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  DBP, Day 1, 24 hour | -1.14 (6.07) | -0.14 (6.24) | -1.14 (6.91) | -0.76 (6.84) | -2.38 (6.05)
  DBP, Day 2, pre-dose: number analyzed (Participants) | 42 | 43 | 43 | 42 | 42
  DBP, Day 2, pre-dose | -1.24 (6.23) | -0.28 (6.08) | -1.02 (6.93) | -0.90 (7.16) | -2.33 (6.43)
  DBP, Day 2, 5 minutes: number analyzed (Participants) | 42 | 43 | 41 | 42 | 42
  DBP, Day 2, 5 minutes | -1.62 (7.05) | -0.81 (5.67) | -0.68 (6.46) | -0.88 (7.27) | -2.62 (5.79)
  DBP, Day 2, 30 minutes: number analyzed (Participants) | 38 | 40 | 38 | 41 | 40
  DBP, Day 2, 30 minutes | -1.71 (6.37) | -0.45 (6.74) | -1.79 (6.99) | -1.80 (6.99) | -2.45 (5.60)
  DBP, Day 2, 1 hour: number analyzed (Participants) | 37 | 40 | 38 | 41 | 40
  DBP, Day 2, 1 hour | -1.65 (7.20) | -0.18 (6.95) | -1.68 (6.87) | -1.10 (6.84) | -1.80 (6.51)
  DBP, Day 8, pre-dose: number analyzed (Participants) | 42 | 43 | 43 | 41 | 39
  DBP, Day 8, pre-dose | -1.50 (8.09) | -1.30 (6.65) | -0.88 (7.49) | 0.02 (6.80) | -2.05 (6.18)
  DBP, Day 8, 5 minutes: number analyzed (Participants) | 42 | 43 | 42 | 41 | 40
  DBP, Day 8, 5 minutes | -2.45 (9.16) | -1.65 (6.94) | -0.98 (7.06) | -0.24 (5.72) | -2.38 (4.86)
  DBP, Day 8, 30 minutes: number analyzed (Participants) | 39 | 40 | 38 | 40 | 38
  DBP, Day 8, 30 minutes | -2.36 (7.19) | -1.93 (6.43) | -1.71 (7.10) | -0.70 (5.89) | -2.58 (4.68)
  DBP, Day 8, 1 hour: number analyzed (Participants) | 38 | 40 | 38 | 40 | 38
  DBP, Day 8, 1 hour | -2.03 (7.15) | -0.93 (6.54) | -1.61 (7.42) | -1.63 (6.95) | -2.16 (5.54)
  DBP, Day 15, pre-dose: number analyzed (Participants) | 43 | 40 | 43 | 41 | 40
  DBP, Day 15, pre-dose | -2.30 (8.17) | -0.10 (7.49) | -1.21 (6.46) | -0.90 (6.81) | -0.63 (6.74)
  DBP, Day 15, 5 minutes: number analyzed (Participants) | 43 | 40 | 42 | 41 | 40
  DBP, Day 15, 5 minutes | -2.70 (8.54) | -0.60 (8.26) | -0.98 (8.15) | -1.85 (6.57) | -1.33 (7.03)
  DBP, Day 15, 30 minutes: number analyzed (Participants) | 39 | 38 | 39 | 41 | 38
  DBP, Day 15, 30 minutes | -3.33 (7.98) | -0.05 (7.15) | -2.15 (7.73) | -2.39 (8.22) | -2.37 (6.26)
  DBP, Day 15, 1 hour: number analyzed (Participants) | 38 | 37 | 39 | 41 | 38
  DBP, Day 15, 1 hour | -3.26 (5.95) | 0.92 (7.57) | -2.23 (7.04) | -2.07 (7.31) | -2.24 (5.51)
  DBP, Day 22, pre-dose: number analyzed (Participants) | 43 | 39 | 43 | 40 | 39
  DBP, Day 22, pre-dose | -1.21 (6.90) | -1.90 (6.53) | -0.67 (6.63) | 0.63 (8.86) | -0.44 (8.08)
  DBP, Day 22, 5 minutes: number analyzed (Participants) | 43 | 39 | 42 | 40 | 39
  DBP, Day 22, 5 minutes | -3.05 (8.91) | -1.62 (6.27) | -1.67 (8.62) | -0.90 (8.44) | -2.54 (7.70)
  DBP, Day 22, 30 minutes: number analyzed (Participants) | 39 | 36 | 39 | 40 | 37
  DBP, Day 22, 30 minutes | -2.51 (7.91) | -2.53 (6.60) | -1.51 (7.44) | -0.98 (8.78) | -1.30 (6.45)
  DBP, Day 22, 1 hour: number analyzed (Participants) | 38 | 36 | 39 | 40 | 37
  DBP, Day 22, 1 hour | -2.89 (6.88) | -1.36 (6.41) | -1.31 (7.16) | -1.35 (8.05) | -2.89 (6.67)
  DBP, Day 27: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  DBP, Day 27 | -2.86 (7.04) | -1.00 (7.53) | -1.43 (6.32) | -0.75 (6.53) | -2.69 (6.22)
  DBP, Day 28, pre-dose: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  DBP, Day 28, pre-dose | -3.67 (6.62) | 0.14 (5.71) | -1.31 (6.66) | 0.25 (8.23) | -1.28 (6.30)
  DBP, Day 28, 15 minutes: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  DBP, Day 28, 15 minutes | -4.37 (7.42) | -1.24 (9.26) | -1.19 (5.58) | -0.63 (8.20) | -1.28 (6.84)
  DBP, Day 28, 30 minutes: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  DBP, Day 28, 30 minutes | -4.37 (7.25) | -0.81 (7.23) | -1.57 (6.01) | -1.05 (8.90) | -2.41 (6.83)
  DBP, Day 28, 1 hour: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  DBP, Day 28, 1 hour | -3.58 (7.11) | -2.00 (6.94) | -1.07 (7.63) | -1.45 (7.37) | -3.62 (5.98)
  DBP, Day 28, 2 hour: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  DBP, Day 28, 2 hour | -4.14 (8.05) | -2.41 (5.89) | -0.93 (6.69) | -2.13 (7.57) | -2.62 (5.42)
  DBP, Day 28, 3 hour: number analyzed (Participants) | 42 | 37 | 42 | 40 | 39
  DBP, Day 28, 3 hour | -3.31 (7.58) | -2.70 (7.08) | -2.71 (5.26) | -2.15 (7.83) | -1.90 (6.18)
  DBP, Day 28, 4 hour: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  DBP, Day 28, 4 hour | -3.30 (7.23) | -1.57 (5.51) | -2.64 (5.92) | -2.10 (7.73) | -2.23 (5.44)
  DBP, Day 28, 8 hour: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  DBP, Day 28, 8 hour | -3.02 (7.16) | -1.03 (5.91) | -1.57 (6.91) | -1.10 (7.73) | -1.33 (6.32)
  DBP, Day 28, 12 hour: number analyzed (Participants) | 43 | 38 | 42 | 40 | 39
  DBP, Day 28, 12 hour | -3.58 (6.27) | -1.82 (6.56) | -1.93 (5.85) | -0.90 (8.45) | -0.97 (6.97)
  DBP, Day 28, 24 hour: number analyzed (Participants) | 43 | 38 | 42 | 40 | 39
  DBP, Day 28, 24 hour | -3.40 (8.66) | -0.71 (7.23) | -2.38 (5.41) | -1.35 (8.34) | -2.21 (6.83)
  DBP, Day 35: number analyzed (Participants) | 43 | 42 | 43 | 41 | 41
  DBP, Day 35 | -2.07 (9.11) | -0.69 (6.38) | -2.33 (8.06) | 0.61 (7.29) | -1.46 (7.02)

5. Primary Outcome: Change From Baseline in Vital Sign Parameter of Heart Rate (HR) Over Time
Description: Vital sign assessment of HR was done at Day 1 (pre-dose, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours and 24 hours post-dose), Day 2 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 8 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 15 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 22 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 27, Day 28 (pre-dose, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours and 24 hours post-dose) and Day 35. A window of plus or minus 5 minutes was allowed during the active treatment visit vital sign assessments. Baseline was defined as the assessment done on Day 1 (pre-dose). The change from Baseline was calculated by subtracting the Baseline value (Day 1, pre-dose) from the individual post-Baseline (Day 1, Day 2, Day 8, Day 15, Day 22, Day 27, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1, pre-dose) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Beats per minute (bpm)
  Day 1, 15 minutes: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 15 minutes | -0.02 (5.82) | 1.02 (5.24) | 0.23 (5.08) | 1.21 (6.32) | 1.60 (4.47)
  Day 1, 30 minutes: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 30 minutes | 0.05 (5.99) | 1.12 (5.55) | 0.47 (6.10) | 1.12 (6.06) | 0.26 (5.40)
  Day 1, 1 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 1 hour | 0.21 (6.16) | 0.33 (5.84) | -0.35 (6.27) | -0.48 (7.19) | 0.43 (4.88)
  Day 1, 2 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 2 hour | -0.23 (5.63) | 0.09 (5.95) | -1.16 (5.63) | -1.19 (5.56) | 0.45 (5.55)
  Day 1, 3 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 3 hour | -0.12 (5.39) | 0.07 (6.25) | -1.19 (6.50) | 0.12 (6.83) | 0.19 (5.71)
  Day 1, 4 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 4 hour | -1.37 (5.94) | -0.53 (6.04) | -0.40 (6.81) | -1.81 (5.64) | 0.05 (6.03)
  Day 1, 8 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 8 hour | -0.70 (6.00) | -0.79 (4.29) | -0.72 (5.15) | -2.14 (5.26) | 0.95 (5.71)
  Day 1, 12 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 12 hour | -1.05 (6.35) | -1.05 (4.77) | -0.72 (6.03) | -1.38 (5.58) | 0.45 (6.66)
  Day 1, 24 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  Day 1, 24 hour | 0.12 (5.49) | -0.40 (5.57) | 0.14 (5.09) | -0.19 (5.06) | 0.64 (5.78)
  Day 2, pre-dose: number analyzed (Participants) | 42 | 43 | 43 | 42 | 42
  Day 2, pre-dose | 0.14 (6.11) | 0.30 (6.06) | 0.14 (5.02) | -0.14 (4.95) | 0.81 (5.61)
  Day 2, 5 minutes: number analyzed (Participants) | 42 | 43 | 41 | 42 | 42
  Day 2, 5 minutes | 1.33 (5.59) | 1.00 (5.81) | -0.12 (5.69) | 0.67 (5.85) | 1.14 (5.34)
  Day 2, 30 minutes: number analyzed (Participants) | 38 | 40 | 38 | 41 | 40
  Day 2, 30 minutes | 0.47 (4.97) | 0.28 (5.80) | -0.08 (6.07) | -0.76 (5.61) | 1.03 (4.70)
  Day 2, 1 hour: number analyzed (Participants) | 37 | 40 | 38 | 41 | 40
  Day 2, 1 hour | -0.38 (4.50) | 0.18 (5.85) | -1.13 (6.63) | -1.29 (6.30) | 1.35 (4.92)
  Day 8, pre-dose: number analyzed (Participants) | 42 | 43 | 43 | 41 | 39
  Day 8, pre-dose | 0.79 (5.72) | -0.84 (6.74) | 1.53 (8.69) | 0.15 (7.80) | 1.36 (6.47)
  Day 8, 5 minutes: number analyzed (Participants) | 42 | 43 | 42 | 41 | 40
  Day 8, 5 minutes | 0.67 (5.15) | -0.56 (6.47) | 1.12 (8.94) | -0.07 (8.13) | 1.85 (6.31)
  Day 8, 30 minutes: number analyzed (Participants) | 39 | 40 | 38 | 40 | 30
  Day 8, 30 minutes | 0.59 (5.92) | -0.15 (6.78) | -1.11 (7.51) | 0.30 (8.46) | 1.66 (5.56)
  Day 8, 1 hour: number analyzed (Participants) | 38 | 40 | 38 | 40 | 38
  Day 8, 1 hour | 0.47 (4.99) | -0.35 (6.91) | -1.26 (6.73) | -0.93 (7.45) | 1.71 (6.23)
  Day 15, pre-dose: number analyzed (Participants) | 43 | 40 | 43 | 41 | 40
  Day 15, pre-dose | -0.35 (7.53) | -0.53 (8.05) | 0.23 (6.79) | -1.10 (8.42) | -0.43 (6.07)
  Day 15, 5 minutes: number analyzed (Participants) | 43 | 40 | 42 | 41 | 40
  Day 15, 5 minutes | -0.05 (6.69) | -0.55 (8.34) | 0.43 (8.14) | -1.17 (8.44) | 0.68 (6.36)
  Day 15, 30 minutes: number analyzed (Participants) | 39 | 38 | 39 | 41 | 38
  Day 15, 30 minutes | -0.72 (6.01) | -0.24 (8.31) | -0.49 (8.42) | -1.68 (8.30) | 0.82 (6.08)
  Day 15, 1 hour: number analyzed (Participants) | 38 | 37 | 39 | 41 | 38
  Day 15, 1 hour | -0.16 (5.25) | -0.81 (7.50) | -1.46 (7.08) | -0.73 (8.33) | 0.13 (5.74)
  Day 22, pre-dose: number analyzed (Participants) | 43 | 39 | 43 | 40 | 39
  Day 22, pre-dose | 0.44 (7.10) | -1.33 (8.21) | 1.33 (7.89) | -0.50 (10.19) | 1.13 (7.45)
  Day 22, 5 minutes: number analyzed (Participants) | 43 | 39 | 42 | 40 | 39
  Day 22, 5 minutes | 0.88 (6.90) | -0.59 (7.27) | 0.88 (8.50) | -0.10 (9.16) | 0.62 (6.74)
  Day 22, 30 minutes: number analyzed (Participants) | 39 | 36 | 39 | 40 | 37
  Day 22, 30 minutes | 0.41 (7.02) | -1.08 (7.69) | 0.05 (8.33) | 0.53 (9.53) | 0.51 (6.42)
  Day 22, 1 hour: number analyzed (Participants) | 38 | 36 | 39 | 40 | 37
  Day 22, 1 hour | -0.21 (6.05) | -1.03 (8.11) | 0.46 (7.45) | 0.28 (9.25) | 0.03 (7.02)
  Day 27: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  Day 27 | -1.70 (6.94) | -1.19 (8.27) | -1.83 (6.58) | -0.75 (8.05) | -0.10 (5.91)
  Day 28, pre-dose: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  Day 28, pre-dose | -1.67 (6.92) | -1.95 (6.99) | -1.26 (5.44) | -0.73 (9.60) | -0.67 (5.89)
  Day 28, 15 minutes: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  Day 28, 15 minutes | -0.67 (7.61) | -1.11 (7.44) | -0.50 (6.95) | -0.03 (10.28) | 0.31 (5.66)
  Day 28, 30 minutes: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 30 minutes | -0.60 (6.97) | -1.84 (6.99) | -0.12 (7.30) | -0.43 (9.47) | 0.26 (5.73)
  Day 28, 1 hour: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 1 hour | -0.44 (6.55) | -1.76 (7.03) | -1.20 (6.75) | -1.18 (9.58) | 0.69 (6.55)
  Day 28, 2 hour: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 2 hour | -1.40 (6.93) | -3.16 (6.13) | -1.20 (6.55) | -0.65 (9.23) | 0.21 (6.88)
  Day 28, 3 hour: number analyzed (Participants) | 42 | 37 | 41 | 40 | 39
  Day 28, 3 hour | -0.55 (6.56) | -1.97 (6.72) | -1.46 (7.41) | -1.53 (8.71) | 0.36 (7.15)
  Day 28, 4 hour: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 4 hour | -0.91 (7.33) | -2.22 (6.94) | -1.24 (6.40) | -1.93 (9.45) | 0.67 (7.19)
  Day 28, 8 hour: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  Day 28, 8 hour | -0.40 (7.47) | -2.14 (6.29) | -1.10 (6.87) | -1.63 (7.88) | 0.05 (7.42)
  Day 28, 12 hour: number analyzed (Participants) | 43 | 38 | 42 | 40 | 39
  Day 28, 12 hour | -1.72 (7.00) | -2.05 (6.15) | -2.02 (7.82) | -0.20 (8.29) | 0.54 (7.57)
  Day 28, 24 hour: number analyzed (Participants) | 43 | 38 | 42 | 40 | 39
  Day 28, 24 hour | -1.58 (7.43) | -1.50 (7.26) | -0.60 (5.49) | -1.33 (7.91) | -0.92 (6.59)
  Day 35: number analyzed (Participants) | 43 | 42 | 43 | 41 | 41
  Day 35 | -0.30 (7.20) | -1.90 (6.80) | -0.56 (6.62) | -3.15 (8.33) | 0.56 (5.96)

6. Primary Outcome: Change From Baseline in Vital Sign Parameter of Respiratory Rate (RR) Over Time
Description: Vital sign assessment of RR was done at Day 1 (pre-dose, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours and 24 hours post-dose), Day 2 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 8 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 15 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 22 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 27, Day 28 (pre-dose, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours and 24 hours post-dose) and Day 35. A window of plus or minus 5 minutes was allowed during the active treatment visit vital sign assessments. Baseline was defined as the assessment done on Day 1 (pre-dose). The change from Baseline was calculated by subtracting the Baseline value (Day 1, pre-dose) from the individual post-Baseline (Day 1, Day 2, Day 8, Day 15, Day 22, Day 27, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1, pre-dose) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Breaths per minute
  Day 1, 15 minutes: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 15 minutes | 0.14 (0.89) | -0.07 (1.12) | -0.16 (1.15) | 0.33 (0.79) | 0.00 (0.99)
  Day 1, 30 minutes: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 30 minutes | 0.07 (1.10) | 0.05 (1.11) | 0.19 (0.96) | 0.96 (1.11) | -0.02 (1.14)
  Day 1, 1 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 1 hour | 0.09 (0.97) | -0.12 (0.96) | -0.23 (1.09) | 0.10 (1.08) | 0.07 (0.97)
  Day 1, 2 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 2 hour | -0.26 (0.93) | 0.19 (1.14) | -0.37 (1.11) | 0.10 (1.05) | 0.21 (1.07)
  Day 1, 3 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 41
  Day 1, 3 hour | -0.02 (0.94) | 0.02 (1.01) | -0.42 (1.10) | 0.31 (1.09) | 0.17 (1.26)
  Day 1, 4 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 4 hour | -0.05 (1.09) | -0.07 (1.01) | -0.12 (1.12) | -0.02 (1.18) | 0.07 (1.11)
  Day 1, 8 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 8 hour | 0.02 (1.20) | -0.02 (0.99) | -0.26 (1.27) | 0.19 (1.09) | 0.07 (0.89)
  Day 1, 12 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 12 hour | -0.14 (1.06) | -0.05 (0.97) | -0.16 (0.92) | 0.24 (1.05) | 0.31 (1.07)
  Day 1, 24 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  Day 1, 24 hour | -0.16 (1.00) | 0.09 (1.25) | -0.45 (0.90) | -0.05 (0.76) | 0.00 (0.83)
  Day 2, pre-dose: number analyzed (Participants) | 42 | 43 | 43 | 42 | 42
  Day 2, pre-dose | 0.00 (0.99) | 0.09 (1.17) | -0.40 (0.90) | -0.02 (0.78) | 0.00 (0.83)
  Day 2, 5 minutes: number analyzed (Participants) | 42 | 43 | 41 | 42 | 42
  Day 2, 5 minutes | 0.29 (0.89) | 0.02 (0.94) | -0.32 (1.01) | 0.10 (1.01) | -0.02 (0.92)
  Day 2, 30 minutes: number analyzed (Participants) | 38 | 40 | 38 | 41 | 40
  Day 2, 30 minutes | 0.18 (1.01) | 0.10 (1.10) | -0.21 (0.93) | -0.15 (1.22) | -0.05 (1.06)
  Day 2, 1 hour: number analyzed (Participants) | 37 | 40 | 38 | 41 | 40
  Day 2, 1 hour | 0.11 (0.97) | 0.13 (1.09) | -0.39 (0.97) | 0.00 (0.74) | 0.10 (0.90)
  Day 8, pre-dose: number analyzed (Participants) | 42 | 43 | 43 | 41 | 39
  Day 8, pre-dose | 0.02 (1.33) | 0.00 (1.00) | -0.37 (1.18) | 0.24 (0.99) | -0.21 (0.95)
  Day 8, 5 minutes: number analyzed (Participants) | 42 | 43 | 42 | 41 | 40
  Day 8, 5 minutes | -0.05 (1.08) | 0.09 (1.00) | -0.43 (1.43) | 0.24 (1.11) | -0.08 (1.07)
  Day 8, 30 minutes: number analyzed (Participants) | 39 | 40 | 38 | 40 | 38
  Day 8, 30 minutes | 0.03 (1.04) | 0.05 (1.32) | -0.50 (1.25) | 0.35 (1.00) | -0.08 (0.97)
  Day 8, 1 hour: number analyzed (Participants) | 38 | 40 | 38 | 40 | 38
  Day 8, 1 hour | 0.05 (1.11) | 0.00 (1.06) | -0.37 (1.15) | 0.08 (1.10) | 0.11 (0.98)
  Day 15, pre-dose: number analyzed (Participants) | 43 | 40 | 43 | 41 | 40
  Day 15, pre-dose | 0.09 (1.15) | -0.05 (1.06) | -0.58 (1.12) | 0.17 (1.09) | 0.00 (0.99)
  Day 15, 5 minutes: number analyzed (Participants) | 43 | 40 | 42 | 41 | 41
  Day 15, 5 minutes | -0.02 (1.24) | -0.15 (1.33) | -0.45 (1.37) | 0.07 (1.10) | -0.08 (1.12)
  Day 15, 30 minutes: number analyzed (Participants) | 39 | 38 | 39 | 41 | 38
  Day 15, 30 minutes | 0.05 (1.15) | -0.08 (1.02) | -0.28 (1.30) | 0.17 (1.32) | 0.03 (1.03)
  Day 15, 1 hour: number analyzed (Participants) | 38 | 37 | 39 | 41 | 38
  Day 15, 1 hour | 0.16 (1.08) | 0.00 (1.37) | -0.64 (1.18) | 0.10 (1.07) | -0.11 (1.01)
  Day 22, pre-dose: number analyzed (Participants) | 43 | 39 | 43 | 40 | 39
  Day 22, pre-dose | -0.02 (1.22) | -0.05 (1.05) | -0.51 (1.18) | 0.10 (1.10) | 0.13 (1.03)
  Day 22, 5 minutes: number analyzed (Participants) | 43 | 39 | 42 | 40 | 39
  Day 22, 5 minutes | 0.07 (1.10) | 0.08 (1.20) | -0.62 (1.45) | 0.25 (1.19) | 0.13 (1.00)
  Day 22, 30 minutes: number analyzed (Participants) | 39 | 36 | 39 | 40 | 37
  Day 22, 30 minutes | 0.10 (1.25) | -0.14 (1.29) | -0.51 (1.00) | 0.20 (1.16) | 0.03 (1.07)
  Day 22, 1 hour: number analyzed (Participants) | 38 | 36 | 39 | 40 | 37
  Day 22, 1 hour | 0.13 (1.19) | 0.11 (1.09) | -0.41 (1.04) | 0.38 (1.17) | 0.00 (1.25)
  Day 27: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  Day 27 | -0.14 (1.06) | 0.11 (0.97) | -0.67 (1.14) | 0.00 (1.28) | 0.26 (1.16)
  Day 28, pre-dose: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  Day 28, pre-dose | -0.09 (1.17) | 0.19 (1.05) | -0.71 (1.20) | 0.10 (1.26) | 0.03 (0.78)
  Day 28, 15 minutes: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 15 minutes | -0.33 (1.23) | -0.08 (1.06) | -0.56 (1.12) | 0.30 (1.36) | -0.05 (1.02)
  Day 28, 30 minutes: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 30 minutes | -0.21 (1.06) | 0.08 (1.23) | -0.32 (1.19) | 0.10 (1.52) | -0.03 (1.04)
  Day 28, 1 hour: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 1 hour | -0.19 (1.30) | -0.08 (1.16) | -0.37 (0.99) | 0.23 (1.54) | -0.05 (1.23)
  Day 28, 2 hour: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 2 hour | -0.33 (1.19) | -0.24 (1.04) | -0.68 (1.21) | 0.30 (1.40) | -0.10 (0.97)
  Day 28, 3 hour: number analyzed (Participants) | 42 | 37 | 41 | 40 | 39
  Day 28, 3 hour | -0.07 (1.30) | 0.00 (1.31) | -0.56 (1.16) | 0.10 (1.37) | -0.13 (1.08)
  Day 28, 4 hour: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 4 hour | -0.05 (1.27) | 0.05 (1.08) | -0.46 (1.14) | 0.25 (1.53) | 0.05 (1.36)
  Day 28, 8 hour: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 8 hour | -0.33 (1.43) | 0.14 (1.00) | -0.54 (0.98) | 0.23 (1.29) | -0.08 (1.18)
  Day 28, 12 hour: number analyzed (Participants) | 43 | 38 | 41 | 40 | 39
  Day 28, 12 hour | -0.35 (1.34) | 0.05 (1.18) | -0.49 (1.14) | 0.20 (1.11) | 0.03 (1.25)
  Day 28, 24 hour: number analyzed (Participants) | 42 | 38 | 42 | 40 | 39
  Day 28, 24 hour | -0.19 (1.19) | -0.03 (0.91) | -0.64 (1.10) | 0.13 (1.45) | -0.18 (1.02)
  Day 35: number analyzed (Participants) | 43 | 42 | 43 | 41 | 41
  Day 35 | -0.35 (1.34) | 0.05 (1.01) | -0.56 (1.10) | 0.07 (1.47) | 0.02 (0.88)

7. Primary Outcome: Change From Baseline in Vital Sign Parameter of Temperature Over Time
Description: Vital sign assessment of temperature was done at Day 1 (pre-dose, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours and 24 hours post-dose), Day 2 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 8 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 15 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 22 (pre-dose, 5 minutes, 30 minutes and 1 hour post-dose), Day 27, Day 28 (pre-dose, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours and 24 hours post-dose) and Day 35. A window of plus or minus 5 minutes was allowed during the active treatment visit vital sign assessments. Baseline was defined as the assessment done on Day 1 (pre-dose). The change from Baseline was calculated by subtracting the Baseline value (Day 1, pre-dose) from the individual post-Baseline (Day 1, Day 2, Day 8, Day 15, Day 22, Day 27, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1, pre-dose) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degree celcius
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Degree celcius
  Day 1, 15 minutes: number analyzed (Participants) | 42 | 43 | 43 | 42 | 42
  Day 1, 15 minutes | 0.03 (0.12) | -0.00 (0.14) | 0.01 (0.11) | 0.04 (0.13) | 0.01 (0.26)
  Day 1, 30 minutes: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 30 minutes | 0.04 (0.21) | -0.01 (0.12) | -0.00 (0.13) | 0.04 (0.12) | 0.03 (0.20)
  Day 1, 1 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 1 hour | 0.05 (0.18) | -0.00 (0.16) | 0.00 (0.13) | 0.04 (0.10) | 0.03 (0.26)
  Day 1, 2 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 2 hour | 0.02 (0.19) | 0.01 (0.20) | 0.02 (0.14) | 0.06 (0.15) | 0.05 (0.21)
  Day 1, 3 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 3 hour | 0.05 (0.20) | -0.00 (0.18) | -0.03 (0.14) | 0.06 (0.16) | 0.01 (0.20)
  Day 1, 4 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 4 hour | 0.05 (0.17) | 0.02 (0.18) | 0.02 (0.18) | 0.05 (0.15) | 0.03 (0.26)
  Day 1, 8 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 8 hour | 0.07 (0.23) | 0.03 (0.20) | 0.03 (0.14) | 0.05 (0.14) | 0.02 (0.20)
  Day 1, 12 hour: number analyzed (Participants) | 43 | 43 | 43 | 42 | 42
  Day 1, 12 hour | 0.12 (0.24) | 0.01 (0.17) | 0.03 (0.18) | 0.05 (0.15) | 0.06 (0.23)
  Day 1, 24 hour: number analyzed (Participants) | 43 | 43 | 44 | 42 | 42
  Day 1, 24 hour | 0.03 (0.16) | -0.03 (0.23) | 0.01 (0.18) | 0.01 (0.19) | 0.00 (0.23)
  Day 2, pre-dose: number analyzed (Participants) | 42 | 43 | 43 | 42 | 42
  Day 2, pre-dose | 0.02 (0.15) | -0.03 (0.23) | 0.02 (0.18) | 0.01 (0.19) | 0.01 (0.23)
  Day 2, 5 minutes: number analyzed (Participants) | 42 | 43 | 41 | 42 | 42
  Day 2, 5 minutes | 0.02 (0.18) | -0.00 (0.18) | 0.01 (0.16) | -0.03 (0.16) | 0.05 (0.21)
  Day 2, 30 minutes: number analyzed (Participants) | 38 | 40 | 38 | 41 | 40
  Day 2, 30 minutes | 0.05 (0.13) | -0.00 (0.15) | -0.01 (0.14) | 0.02 (0.17) | 0.06 (0.22)
  Day 2, 1 hour: number analyzed (Participants) | 37 | 40 | 38 | 41 | 40
  Day 2, 1 hour | 0.04 (0.11) | -0.00 (0.16) | -0.00 (0.16) | 0.03 (0.14) | 0.04 (0.23)
  Day 8, pre-dose: number analyzed (Participants) | 42 | 43 | 43 | 41 | 39
  Day 8, pre-dose | 0.07 (0.25) | 0.03 (0.17) | 0.00 (0.24) | 0.02 (0.18) | -0.01 (0.22)
  Day 8, 5 minutes: number analyzed (Participants) | 42 | 43 | 42 | 41 | 40
  Day 8, 5 minutes | 0.05 (0.21) | 0.03 (0.18) | 0.01 (0.19) | 0.01 (0.17) | 0.03 (0.21)
  Day 8, 30 minutes: number analyzed (Participants) | 39 | 40 | 38 | 40 | 38
  Day 8, 30 minutes | 0.06 (0.20) | 0.00 (0.16) | -0.03 (0.19) | 0.03 (0.17) | 0.04 (0.20)
  Day 8, 1 hour: number analyzed (Participants) | 38 | 40 | 38 | 40 | 38
  Day 8, 1 hour | 0.03 (0.14) | 0.01 (0.16) | -0.02 (0.21) | 0.03 (0.20) | 0.03 (0.24)
  Day 15, pre-dose: number analyzed (Participants) | 43 | 40 | 43 | 41 | 40
  Day 15, pre-dose | 0.03 (0.24) | 0.00 (0.17) | 0.02 (0.19) | 0.06 (0.21) | 0.01 (0.19)
  Day 15, 5 minutes: number analyzed (Participants) | 43 | 40 | 42 | 41 | 40
  Day 15, 5 minutes | 0.05 (0.20) | 0.01 (0.18) | 0.01 (0.20) | 0.05 (0.17) | 0.02 (0.24)
  Day 15, 30 minutes: number analyzed (Participants) | 39 | 38 | 39 | 41 | 38
  Day 15, 30 minutes | 0.07 (0.20) | -0.01 (0.20) | -0.01 (0.18) | 0.05 (0.18) | 0.03 (0.21)
  Day 15, 1 hour: number analyzed (Participants) | 38 | 37 | 39 | 41 | 38
  Day 15, 1 hour | 0.05 (0.14) | 0.04 (0.15) | -0.02 (0.19) | 0.04 (0.15) | 0.01 (0.15)
  Day 22, pre-dose: number analyzed (Participants) | 43 | 39 | 43 | 40 | 39
  Day 22, pre-dose | 0.00 (0.20) | 0.04 (0.25) | -0.02 (0.13) | -0.01 (0.25) | 0.01 (0.10)
  Day 22, 5 minutes: number analyzed (Participants) | 43 | 39 | 42 | 40 | 39
  Day 22, 5 minutes | 0.01 (0.17) | 0.04 (0.23) | -0.00 (0.16) | -0.01 (0.20) | 0.00 (0.12)
  Day 22, 30 minutes: number analyzed (Participants) | 39 | 36 | 39 | 40 | 37
  Day 22, 30 minutes | 0.04 (0.16) | 0.04 (0.21) | -0.03 (0.12) | 0.03 (0.23) | 0.01 (0.10)
  Day 22, 1 hour: number analyzed (Participants) | 38 | 36 | 39 | 40 | 37
  Day 22, 1 hour | 0.02 (0.17) | 0.05 (0.21) | 0.01 (0.14) | 0.02 (0.22) | 0.01 (0.09)
  Day 27: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  Day 27 | 0.04 (0.21) | 0.01 (0.24) | 0.01 (0.20) | 0.05 (0.21) | 0.03 (0.13)
  Day 28, pre-dose: number analyzed (Participants) | 43 | 37 | 42 | 40 | 39
  Day 28, pre-dose | -0.00 (0.17) | -0.00 (0.18) | -0.01 (0.19) | 0.00 (0.19) | -0.01 (0.18)
  Day 28, 15 minutes: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 15 minutes | 0.02 (0.17) | -0.00 (0.20) | 0.00 (0.18) | 0.04 (0.21) | -0.00 (0.17)
  Day 28, 30 minutes: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 30 minutes | 0.02 (0.15) | -0.01 (0.24) | -0.01 (0.17) | 0.05 (0.24) | 0.02 (0.17)
  Day 28, 1 hour: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 1 hour | 0.02 (0.17) | -0.04 (0.28) | -0.01 (0.15) | 0.04 (0.24) | 0.00 (0.12)
  Day 28, 2 hour: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 2 hour | 0.03 (0.19) | -0.00 (0.25) | -0.04 (0.16) | 0.04 (0.18) | 0.02 (0.13)
  Day 28, 3 hour: number analyzed (Participants) | 42 | 37 | 41 | 40 | 39
  Day 28, 3 hour | 0.02 (0.13) | 0.01 (0.26) | -0.01 (0.21) | 0.02 (0.22) | 0.00 (0.16)
  Day 28, 4 hour: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 4 hour | -0.01 (0.25) | 0.00 (0.27) | -0.02 (0.16) | 0.02 (0.22) | 0.01 (0.11)
  Day 28, 8 hour: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28, 8 hour | 0.05 (0.21) | 0.05 (0.24) | 0.00 (0.17) | 0.05 (0.17) | 0.02 (0.16)
  Day 28, 12 hour: number analyzed (Participants) | 42 | 38 | 41 | 40 | 39
  Day 28, 12 hour | 0.05 (0.16) | 0.06 (0.27) | 0.01 (0.18) | 0.05 (0.21) | -0.01 (0.15)
  Day 28, 24 hour: number analyzed (Participants) | 43 | 38 | 42 | 40 | 39
  Day 28, 24 hour | -0.01 (0.22) | -0.02 (0.25) | -0.09 (0.35) | 0.02 (0.26) | -0.02 (0.19)
  Day 35: number analyzed (Participants) | 43 | 42 | 43 | 41 | 41
  Day 35 | -0.00 (0.24) | 0.07 (0.18) | -0.02 (0.18) | 0.07 (0.23) | 0.02 (0.32)

8. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Values Over Time
Description: 12-lead ECG was obtained in the rested state. Participants lied in supine position with ECG leads on for at least 5 minutes prior to ECG recording. The ECG was performed at Day 1 (pre-dose and post-dose), Day 8, Day 15, Day 22, Day 28 (pre-dose and pre-dose) and Day 35, and included the assessment of PR interval, QRS interval, QT interval and QTc interval. Baseline was defined as the assessment done on Day 1 (pre-dose). The change from Baseline was calculated by subtracting the Baseline value (Day 1, pre-dose) from the individual post-Baseline (Day 1 [post-dose], Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1, pre-dose) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Millisecond
  PR interval, Day 1, post-dose: number analyzed (Participants) | 42 | 43 | 43 | 41 | 42
  PR interval, Day 1, post-dose | 0.12 (9.92) | 1.47 (13.07) | 0.58 (12.43) | 0.32 (9.96) | 1.57 (11.91)
  PR interval, Day 8: number analyzed (Participants) | 42 | 43 | 42 | 41 | 40
  PR interval, Day 8 | -0.26 (17.29) | -3.42 (18.04) | 0.45 (14.15) | -2.46 (14.66) | -3.63 (15.56)
  PR interval, Day 15: number analyzed (Participants) | 42 | 40 | 41 | 41 | 40
  PR interval, Day 15 | -5.79 (15.29) | -3.20 (16.45) | -5.10 (19.64) | -0.78 (12.10) | -1.03 (12.96)
  PR interval, Day 22: number analyzed (Participants) | 42 | 39 | 42 | 40 | 39
  PR interval, Day 22 | -2.38 (16.84) | -0.31 (18.12) | -1.19 (14.86) | 0.15 (12.31) | -1.46 (14.71)
  PR interval, Day 28, pre-dose: number analyzed (Participants) | 42 | 37 | 41 | 40 | 39
  PR interval, Day 28, pre-dose | -0.55 (14.81) | -3.46 (18.59) | -2.39 (14.43) | 3.70 (13.45) | 0.31 (17.74)
  PR interval, Day 28, post-dose: number analyzed (Participants) | 42 | 37 | 41 | 40 | 39
  PR interval, Day 28, post-dose | -1.98 (15.72) | -1.22 (17.40) | -1.59 (16.55) | 1.88 (15.35) | 3.33 (13.27)
  PR interval, Day 35: number analyzed (Participants) | 42 | 41 | 42 | 41 | 41
  PR interval, Day 35 | -0.07 (16.43) | -1.22 (25.54) | 0.48 (19.88) | 1.95 (13.81) | 1.15 (10.41)
  QRS interval, Day 1, post-dose: number analyzed (Participants) | 42 | 43 | 43 | 41 | 42
  QRS interval, Day 1, post-dose | -0.83 (8.31) | 1.07 (9.67) | -0.16 (3.31) | 0.54 (7.18) | 1.45 (8.12)
  QRS interval, Day 8: number analyzed (Participants) | 42 | 43 | 42 | 41 | 40
  QRS interval, Day 8 | -0.50 (7.74) | -17.49 (107.04) | 0.81 (6.78) | 0.56 (7.23) | 0.85 (10.15)
  QRS interval, Day 15: number analyzed (Participants) | 42 | 40 | 41 | 41 | 40
  QRS interval, Day 15 | -1.05 (6.89) | -16.15 (110.73) | -0.17 (6.26) | -1.37 (11.87) | 0.80 (8.16)
  QRS interval, Day 22: number analyzed (Participants) | 42 | 39 | 42 | 40 | 39
  QRS interval, Day 22 | 0.14 (5.88) | -19.31 (112.93) | -0.26 (7.15) | -1.00 (5.43) | 0.28 (9.51)
  QRS interval, Day 28, pre-dose: number analyzed (Participants) | 42 | 37 | 41 | 40 | 39
  QRS interval, Day 28, pre-dose | -0.81 (9.55) | -20.00 (120.11) | -0.54 (6.24) | -1.28 (6.80) | -0.54 (7.41)
  QRS interval, Day 28, post-dose: number analyzed (Participants) | 42 | 37 | 41 | 40 | 39
  QRS interval, Day 28, post-dose | -0.14 (11.71) | -19.38 (120.28) | -0.85 (7.62) | -0.03 (6.62) | 0.21 (9.09)
  QRS interval, Day 35: number analyzed (Participants) | 42 | 41 | 42 | 41 | 41
  QRS interval, Day 35 | -0.36 (6.55) | -12.39 (112.59) | -1.21 (5.58) | -1.17 (10.59) | 0.83 (8.89)
  QT interval, Day 1, post-dose: number analyzed (Participants) | 42 | 43 | 43 | 41 | 42
  QT interval, Day 1, post-dose | -0.29 (14.09) | -2.44 (20.72) | 1.23 (18.96) | 3.49 (18.44) | 1.17 (17.14)
  QT interval, Day 8: number analyzed (Participants) | 42 | 43 | 42 | 41 | 40
  QT interval, Day 8 | -1.17 (18.65) | -7.56 (32.44) | -2.74 (21.35) | 0.68 (13.49) | -2.98 (25.80)
  QT interval, Day 15: number analyzed (Participants) | 42 | 40 | 41 | 41 | 40
  QT interval, Day 15 | 0.93 (23.43) | 0.40 (21.66) | -0.66 (22.63) | -0.98 (15.75) | 1.53 (19.98)
  QT interval, Day 22: number analyzed (Participants) | 42 | 39 | 42 | 40 | 39
  QT interval, Day 22 | 1.38 (20.93) | 1.31 (21.31) | 1.36 (22.41) | -6.00 (18.92) | 0.64 (18.54)
  QT interval, Day 28, pre-dose: number analyzed (Participants) | 42 | 37 | 41 | 40 | 39
  QT interval, Day 28, pre-dose | 9.17 (25.76) | 1.62 (19.05) | 1.46 (27.63) | 3.48 (20.88) | 1.00 (18.20)
  QT interval, Day 28, post-dose: number analyzed (Participants) | 42 | 37 | 41 | 40 | 39
  QT interval, Day 28, post-dose | 0.90 (34.52) | 4.27 (18.31) | 3.80 (24.89) | 4.35 (24.70) | -1.28 (24.60)
  QT interval, Day 35: number analyzed (Participants) | 42 | 41 | 42 | 41 | 41
  QT interval, Day 35 | 2.10 (22.76) | 4.56 (22.44) | 0.36 (20.27) | 5.12 (26.01) | 4.27 (27.43)
  QTc interval, Day 1, post-dose: number analyzed (Participants) | 42 | 43 | 43 | 41 | 42
  QTc interval, Day 1, post-dose | -2.52 (16.05) | -1.60 (16.31) | 1.28 (14.46) | 3.37 (18.91) | -1.71 (23.06)
  QTc interval, Day 8: number analyzed (Participants) | 42 | 43 | 42 | 41 | 40
  QTc interval, Day 8 | 5.02 (21.98) | -3.40 (27.38) | 3.64 (20.77) | 4.17 (20.65) | 1.45 (25.90)
  QTc interval, Day 15: number analyzed (Participants) | 42 | 40 | 41 | 41 | 40
  QTc interval, Day 15 | -0.57 (21.03) | -3.05 (26.25) | 2.78 (15.96) | 0.68 (19.64) | 4.40 (23.37)
  QTc interval, Day 22: number analyzed (Participants) | 42 | 39 | 42 | 40 | 39
  QTc interval, Day 22 | 3.21 (17.87) | -4.21 (17.59) | 5.52 (17.55) | -4.13 (23.18) | -0.10 (22.32)
  QTc interval, Day 28, pre-dose: number analyzed (Participants) | 42 | 37 | 41 | 40 | 39
  QTc interval, Day 28, pre-dose | 4.98 (17.02) | 2.35 (18.90) | -0.71 (24.18) | 1.50 (19.86) | -4.67 (19.30)
  QTc interval, Day 28, post-dose: number analyzed (Participants) | 42 | 37 | 41 | 40 | 39
  QTc interval, Day 28, post-dose | 2.05 (21.32) | 0.54 (21.20) | 2.39 (23.09) | 0.83 (19.86) | -4.44 (20.43)
  QTc interval, Day 35: number analyzed (Participants) | 42 | 41 | 42 | 41 | 41
  QTc interval, Day 35 | 2.38 (19.88) | -0.05 (21.78) | 2.90 (16.15) | 0.63 (26.55) | -1.34 (28.57)

9. Primary Outcome: Change From Baseline in Hematology Parameters of Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet and White Blood Cell (WBC) Count Over Time
Description: Assessment for basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelet and white blood cell (WBC) count were performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Giga cells per liter
  Baseophil count, Day 8: number analyzed (Participants) | 36 | 35 | 36 | 31 | 37
  Baseophil count, Day 8 | 0.01 (0.02) | 0.00 (0.02) | 0.00 (0.01) | 0.00 (0.02) | -0.00 (0.02)
  Baseophil count, Day 15: number analyzed (Participants) | 38 | 32 | 35 | 33 | 38
  Baseophil count, Day 15 | 0.01 (0.02) | 0.01 (0.03) | 0.01 (0.03) | -0.00 (0.02) | -0.00 (0.02)
  Baseophil count, Day 22: number analyzed (Participants) | 34 | 33 | 37 | 35 | 38
  Baseophil count, Day 22 | 0.01 (0.01) | 0.01 (0.03) | -0.00 (0.02) | -0.00 (0.02) | -0.01 (0.02)
  Baseophil count, Day 28: number analyzed (Participants) | 37 | 29 | 35 | 32 | 39
  Baseophil count, Day 28 | 0.01 (0.02) | 0.00 (0.02) | 0.00 (0.02) | -0.00 (0.02) | -0.00 (0.02)
  Baseophil count Day 35: number analyzed (Participants) | 36 | 32 | 37 | 33 | 37
  Baseophil count Day 35 | 0.00 (0.02) | 0.01 (0.02) | 0.00 (0.02) | 0.00 (0.02) | -0.00 (0.02)
  Eosinophil count, Day 8: number analyzed (Participants) | 36 | 35 | 36 | 31 | 37
  Eosinophil count, Day 8 | 0.01 (0.14) | 0.01 (0.13) | 0.03 (0.17) | -0.01 (0.09) | 0.01 (0.14)
  Eosinophil count, Day 15: number analyzed (Participants) | 38 | 32 | 35 | 33 | 38
  Eosinophil count, Day 15 | -0.04 (0.13) | 0.01 (0.12) | 0.04 (0.28) | 0.01 (0.11) | -0.03 (0.12)
  Eosinophil count, Day 22: number analyzed (Participants) | 34 | 33 | 37 | 35 | 38
  Eosinophil count, Day 22 | -0.01 (0.21) | 0.01 (0.10) | 0.01 (0.15) | 0.02 (0.20) | 0.03 (0.16)
  Eosinophil count, Day 28: number analyzed (Participants) | 37 | 29 | 35 | 32 | 39
  Eosinophil count, Day 28 | -0.05 (0.11) | 0.02 (0.13) | 0.02 (0.27) | -0.00 (0.10) | 0.02 (0.17)
  Eosinophil count, Day 35: number analyzed (Participants) | 36 | 32 | 37 | 33 | 37
  Eosinophil count, Day 35 | -0.02 (0.15) | -0.01 (0.14) | 0.03 (0.24) | -0.02 (0.11) | 0.05 (0.21)
  Lymphocyte count, Day 8: number analyzed (Participants) | 36 | 35 | 36 | 31 | 37
  Lymphocyte count, Day 8 | 0.12 (0.44) | 0.20 (0.59) | 0.10 (0.46) | 0.12 (0.53) | 0.20 (0.58)
  Lymphocyte count, Day 15: number analyzed (Participants) | 38 | 32 | 35 | 33 | 38
  Lymphocyte count, Day 15 | 0.22 (0.52) | 0.10 (0.58) | 0.16 (0.41) | 0.11 (0.46) | 0.05 (0.46)
  Lymphocyte count, Day 22: number analyzed (Participants) | 34 | 33 | 37 | 35 | 38
  Lymphocyte count, Day 22 | 0.14 (0.46) | 0.17 (0.54) | 0.22 (0.43) | -0.00 (0.43) | 0.04 (0.36)
  Lymphocyte count, Day 28: number analyzed (Participants) | 37 | 29 | 35 | 32 | 39
  Lymphocyte count, Day 28 | 0.05 (0.48) | -0.03 (0.49) | 0.49 (0.47) | -0.02 (0.47) | -0.07 (0.47)
  Lymphocyte count, Day 35: number analyzed (Participants) | 36 | 32 | 37 | 33 | 37
  Lymphocyte count, Day 35 | 0.16 (0.45) | 0.15 (0.58) | 0.18 (0.43) | 0.06 (0.46) | 0.10 (0.57)
  Monocyte count, Day 8: number analyzed (Participants) | 36 | 35 | 36 | 31 | 37
  Monocyte count, Day 8 | 0.04 (0.11) | 0.02 (0.16) | 0.03 (0.13) | 0.04 (0.15) | 0.05 (0.18)
  Monocyte count, Day 15: number analyzed (Participants) | 38 | 32 | 35 | 33 | 38
  Monocyte count, Day 15 | 0.02 (0.12) | 0.02 (0.18) | 0.04 (0.12) | 0.04 (0.14) | 0.04 (0.15)
  Monocyte count, Day 22: number analyzed (Participants) | 34 | 33 | 37 | 35 | 38
  Monocyte count, Day 22 | 0.05 (0.13) | 0.05 (0.19) | 0.01 (0.13) | 0.00 (0.18) | 0.05 (0.16)
  Monocyte count, Day 28: number analyzed (Participants) | 37 | 29 | 35 | 32 | 39
  Monocyte count, Day 28 | 0.00 (0.11) | -0.03 (0.15) | -0.00 (0.13) | -0.01 (0.11) | 0.00 (0.17)
  Monocyte count, Day 35: number analyzed (Participants) | 36 | 32 | 37 | 33 | 37
  Monocyte count, Day 35 | 0.03 (0.11) | 0.02 (0.15) | 0.00 (0.15) | -0.01 (0.15) | 0.02 (0.16)
  Neutrophil count, Day 8: number analyzed (Participants) | 36 | 35 | 36 | 31 | 37
  Neutrophil count, Day 8 | 0.01 (1.08) | 0.37 (1.29) | 0.11 (1.05) | 0.10 (1.23) | 0.03 (1.11)
  Neutrophil count, Day 15: number analyzed (Participants) | 38 | 32 | 35 | 33 | 38
  Neutrophil count, Day 15 | 0.15 (0.83) | 0.55 (1.19) | 0.27 (0.88) | 0.31 (1.27) | 0.46 (1.40)
  Neutrophil count, Day 22: number analyzed (Participants) | 34 | 33 | 37 | 35 | 38
  Neutrophil count, Day 22 | -0.07 (0.82) | 0.56 (1.31) | 0.31 (0.71) | 0.14 (1.38) | 0.20 (1.59)
  Neutrophil count, Day 28: number analyzed (Participants) | 37 | 29 | 35 | 32 | 39
  Neutrophil count, Day 28 | 0.08 (1.34) | 0.35 (1.23) | -0.18 (0.96) | 0.19 (1.21) | 0.26 (1.28)
  Neutrophil count, Day 35: number analyzed (Participants) | 36 | 32 | 37 | 33 | 37
  Neutrophil count, Day 35 | 0.05 (1.27) | 0.29 (1.18) | 0.09 (0.63) | 0.28 (1.13) | 0.55 (1.40)
  Platelet count, Day 8: number analyzed (Participants) | 38 | 37 | 38 | 37 | 40
  Platelet count, Day 8 | 6.37 (35.76) | 4.03 (40.19) | 2.34 (26.94) | 12.14 (28.82) | 5.75 (23.95)
  Platelet count, Day 15: number analyzed (Participants) | 36 | 33 | 39 | 35 | 40
  Platelet count, Day 15 | 15.19 (41.90) | 13.45 (39.23) | 13.10 (28.86) | 15.40 (30.99) | 7.73 (28.91)
  Platelet count, Day 22: number analyzed (Participants) | 36 | 35 | 38 | 37 | 39
  Platelet count, Day 22 | 9.28 (33.79) | 9.49 (42.29) | 16.42 (27.73) | 19.70 (29.51) | 4.49 (30.38)
  Platelet count, Day 28: number analyzed (Participants) | 39 | 32 | 38 | 37 | 40
  Platelet count, Day 28 | -3.05 (33.65) | 3.81 (45.00) | 7.11 (21.05) | 5.22 (34.65) | 8.73 (43.33)
  Platelet count, Day 35: number analyzed (Participants) | 35 | 37 | 40 | 34 | 40
  Platelet count, Day 35 | 10.89 (31.69) | 6.27 (42.88) | 11.58 (26.85) | 20.65 (35.89) | 15.75 (37.58)
  WBC count, Day 8: number analyzed (Participants) | 39 | 41 | 38 | 38 | 41
  WBC count, Day 8 | 0.15 (1.36) | 0.43 (1.66) | 0.37 (1.27) | 0.09 (1.45) | 0.22 (1.49)
  WBC count, Day 15: number analyzed (Participants) | 39 | 35 | 39 | 36 | 40
  WBC count, Day 15 | 0.35 (0.94) | 0.67 (1.36) | 0.59 (1.10) | 0.44 (1.33) | 0.49 (1.60)
  WBC count, Day 22: number analyzed (Participants) | 38 | 37 | 39 | 38 | 39
  WBC count, Day 22 | 0.15 (0.92) | 0.75 (1.64) | 0.58 (0.94) | 0.18 (1.62) | 0.31 (1.76)
  WBC count, Day 28: number analyzed (Participants) | 40 | 34 | 39 | 38 | 40
  WBC count, Day 28 | 0.12 (1.43) | 0.21 (1.56) | 0.03 (1.20) | 0.02 (1.41) | 0.20 (1.46)
  WBC count, Day 35: number analyzed (Participants) | 36 | 39 | 40 | 36 | 40
  WBC count, Day 35 | 0.23 (1.29) | 0.29 (1.53) | 0.34 (0.90) | 0.26 (1.21) | 0.66 (1.68)

10. Primary Outcome: Change From Baseline in Hematology Parameter of Red Blood Cell (RBC) Count Over Time
Description: Assessment for RBC count was performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Trillion cells per liter
  Day 8: number analyzed (Participants) | 40 | 41 | 40 | 38 | 41
  Day 8 | -0.02 (0.19) | 0.03 (0.31) | -0.02 (0.24) | 0.03 (0.23) | 0.03 (0.20)
  Day 15: number analyzed (Participants) | 39 | 35 | 41 | 36 | 40
  Day 15 | 0.01 (0.19) | 0.02 (0.39) | -0.04 (0.22) | -0.03 (0.21) | 0.02 (0.24)
  Day 22: number analyzed (Participants) | 38 | 37 | 42 | 38 | 39
  Day 22 | 0.04 (0.48) | 0.03 (0.36) | -0.04 (0.22) | -0.01 (0.27) | -0.01 (0.20)
  Day 28: number analyzed (Participants) | 40 | 35 | 41 | 38 | 40
  Day 28 | -0.02 (0.25) | -0.10 (0.38) | -0.11 (0.23) | -0.09 (0.33) | -0.12 (0.23)
  Day 35: number analyzed (Participants) | 36 | 39 | 42 | 36 | 40
  Day 35 | -0.08 (0.27) | -0.10 (0.35) | -0.14 (0.21) | -0.13 (0.41) | -0.12 (0.21)

11. Primary Outcome: Change From Baseline in Hematology Parameter of Hematocrit Over Time
Description: Assessment for hematocrit was performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Ratio
  Day 8: number analyzed (Participants) | 35 | 36 | 39 | 36 | 30
  Day 8 | -0.00 (0.02) | 0.00 (0.03) | -0.00 (0.03) | 0.00 (0.03) | 0.00 (0.02)
  Day 15: number analyzed (Participants) | 34 | 32 | 37 | 32 | 32
  Day 15 | 0.00 (0.02) | 0.00 (0.04) | -0.00 (0.02) | -0.00 (0.02) | -0.00 (0.02)
  Day 22: number analyzed (Participants) | 35 | 32 | 40 | 35 | 32
  Day 22 | 0.01 (0.05) | 0.01 (0.03) | -0.00 (0.02) | -0.00 (0.03) | -0.00 (0.02)
  Day 28: number analyzed (Participants) | 32 | 27 | 34 | 34 | 27
  Day 28 | -0.00 (0.02) | -0.01 (0.04) | -0.01 (0.02) | -0.01 (0.04) | -0.01 (0.03)
  Day 35: number analyzed (Participants) | 34 | 31 | 37 | 31 | 26
  Day 35 | -0.00 (0.03) | -0.01 (0.03) | -0.01 (0.02) | -0.01 (0.03) | -0.01 (0.02)

12. Primary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin Over Time
Description: Assessment for hemoglobin was performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Gram per liter
  Day 8: number analyzed (Participants) | 40 | 41 | 40 | 38 | 41
  Day 8 | -0.75 (5.17) | 1.49 (9.28) | -0.03 (7.36) | 0.47 (8.03) | 1.44 (6.58)
  Day 15: number analyzed (Participants) | 39 | 35 | 41 | 36 | 40
  Day 15 | 0.31 (5.13) | 1.09 (11.65) | -0.32 (7.21) | -0.81 (8.25) | 0.40 (6.70)
  Day 22: number analyzed (Participants) | 38 | 37 | 42 | 38 | 39
  Day 22 | -1.08 (5.87) | 1.05 (10.71) | -0.57 (7.56) | -0.82 (9.70) | -0.05 (5.92)
  Day 28: number analyzed (Participants) | 40 | 35 | 41 | 38 | 40
  Day 28 | -0.43 (7.34) | -2.60 (11.34) | -2.32 (7.83) | -2.58 (10.49) | -3.83 (6.88)
  Day 35: number analyzed (Participants) | 36 | 39 | 42 | 36 | 40
  Day 35 | -2.19 (8.37) | -2.33 (11.10) | -3.50 (7.53) | -4.75 (9.87) | -3.08 (6.16)

13. Primary Outcome: Change From Baseline in Hematology Parameter of Mean Corpuscular Hemoglobin Over Time
Description: Assessment for mean corpuscular hemoglobin was performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picogram per cell
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Picogram per cell
  Day 8: number analyzed (Participants) | 40 | 41 | 40 | 38 | 41
  Day 8 | 0.00 (0.72) | 0.15 (0.79) | 0.23 (0.62) | -0.16 (0.82) | 0.17 (0.67)
  Day 15: number analyzed (Participants) | 39 | 35 | 41 | 36 | 40
  Day 15 | 0.03 (0.58) | 0.23 (1.14) | 0.27 (0.63) | -0.03 (0.81) | -0.08 (0.53)
  Day 22: number analyzed (Participants) | 38 | 37 | 42 | 38 | 39
  Day 22 | -0.24 (1.79) | 0.14 (0.79) | 0.14 (0.65) | -0.18 (0.90) | 0.10 (0.64)
  Day 28: number analyzed (Participants) | 40 | 35 | 41 | 38 | 40
  Day 28 | 0.10 (0.74) | 0.11 (0.96) | 0.39 (0.67) | 0.03 (0.94) | 0.00 (0.60)
  Day 35: number analyzed (Participants) | 36 | 39 | 42 | 36 | 40
  Day 35 | 0.11 (0.82) | 0.05 (1.36) | 0.38 (0.66) | -0.11 (1.74) | 0.08 (0.73)

14. Primary Outcome: Change From Baseline in Hematology Parameter of Mean Corpuscular Hemoglobin Concentration Over Time
Description: Assessment for mean corpuscular hemoglobin concentration was performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram hemoglobin per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Gram hemoglobin per liter
  Day 8: number analyzed (Participants) | 35 | 36 | 39 | 36 | 30
  Day 8 | -1.43 (8.10) | 0.00 (7.56) | 0.77 (8.39) | 0.56 (9.24) | 3.33 (9.24)
  Day 15: number analyzed (Participants) | 34 | 32 | 37 | 32 | 32
  Day 15 | 0.59 (7.36) | 0.31 (8.22) | 2.16 (7.50) | -0.63 (11.34) | 0.31 (8.61)
  Day 22: number analyzed (Participants) | 35 | 32 | 40 | 35 | 32
  Day 22 | -4.00 (21.58) | -1.25 (8.33) | 0.25 (9.47) | -2.29 (11.65) | 1.56 (7.67)
  Day 28: number analyzed (Participants) | 32 | 27 | 34 | 34 | 27
  Day 28 | -1.56 (8.08) | 1.85 (8.34) | 1.47 (6.57) | -0.59 (12.78) | 0.00 (8.77)
  Day 35: number analyzed (Participants) | 34 | 31 | 37 | 31 | 26
  Day 35 | -2.35 (7.81) | 0.32 (11.69) | -0.81 (7.22) | 0.32 (12.51) | -1.54 (7.32)

15. Primary Outcome: Change From Baseline in Hematology Parameter of Mean Corpuscular Volume Over Time
Description: Assessment for mean corpuscular volume was performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Femtoliter
  Day 8: number analyzed (Participants) | 35 | 36 | 39 | 36 | 30
  Day 8 | 0.20 (1.21) | 0.28 (1.77) | 0.18 (1.68) | -0.33 (2.24) | -0.17 (1.53)
  Day 15: number analyzed (Participants) | 34 | 32 | 37 | 32 | 32
  Day 15 | 0.29 (1.29) | 0.69 (3.35) | 0.11 (1.54) | -0.06 (2.71) | -0.03 (1.45)
  Day 22: number analyzed (Participants) | 35 | 32 | 40 | 35 | 32
  Day 22 | 0.17 (1.98) | 0.59 (1.70) | 0.05 (1.72) | 0.03 (2.27) | 0.13 (1.66)
  Day 28: number analyzed (Participants) | 32 | 27 | 34 | 34 | 27
  Day 28 | 0.81 (1.89) | -0.19 (2.43) | 0.29 (1.17) | 0.29 (2.70) | 0.22 (1.72)
  Day 35: number analyzed (Participants) | 34 | 31 | 37 | 31 | 26
  Day 35 | 1.00 (1.74) | 0.74 (3.01) | 0.73 (1.63) | -0.71 (4.27) | 0.77 (1.70)

16. Primary Outcome: Change From Baseline in Coagulation Parameters of Activated Partial Thromplastin Time (aPTT) and Prothrombin Time (PT) Over Time
Description: Assessment for aPTT and PT were performed on Day 1, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 28 and Day 35) values.
Time Frame: Baseline (Day 1), Day 28 and Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Seconds
  aPTT, Day 28: number analyzed (Participants) | 33 | 35 | 31 | 33 | 34
  aPTT, Day 28 | 0.53 (6.78) | 1.51 (9.88) | -1.58 (6.98) | 1.41 (13.03) | 1.26 (10.07)
  aPTT, Day 35: number analyzed (Participants) | 34 | 38 | 33 | 37 | 33
  aPTT, Day 35 | -0.43 (6.99) | -1.73 (4.28) | -1.46 (4.31) | -1.28 (4.33) | -0.84 (5.26)
  PT, Day 28: number analyzed (Participants) | 34 | 34 | 31 | 33 | 35
  PT, Day 28 | -0.28 (1.62) | 0.18 (2.68) | 0.20 (2.99) | -0.18 (1.43) | -0.36 (1.99)
  PT, Day 35: number analyzed (Participants) | 35 | 37 | 33 | 37 | 33
  PT, Day 35 | -0.49 (1.62) | -0.45 (1.13) | -0.26 (0.83) | -0.47 (2.07) | -0.44 (0.94)

17. Primary Outcome: Change From Baseline in Coagulation Parameter of International Normalized Ratio Over Time
Description: Assessment for international normalized ratio was performed on Day 1, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 28 and Day 35) values.
Time Frame: Baseline (Day 1), Day 28 and Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Ratio
  Day 28: number analyzed (Participants) | 34 | 34 | 31 | 33 | 25
  Day 28 | -0.02 (0.13) | 0.02 (0.24) | 0.01 (0.24) | -0.01 (0.11) | -0.03 (0.16)
  Day 35: number analyzed (Participants) | 35 | 37 | 33 | 37 | 33
  Day 35 | -0.04 (0.13) | -0.03 (0.09) | -0.02 (0.07) | -0.04 (0.16) | -0.04 (0.07)

18. Primary Outcome: Change From Baseline in Chemistry Parameters of Alanine Aminotransferase (ALT), Aspartate Aminotrasferase (AST), Alkaline Phosphatase (ALP), Creatinine Phosphokinase and Lactate Dehydrogenase (LDH) Over Time
Description: Assessment for ALT, AST, ALP, creatinine phosphokinase and LDH were performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
International units per liter
  ALT, Day 8: number analyzed (Participants) | 39 | 40 | 38 | 34 | 39
  ALT, Day 8 | 0.90 (8.33) | -0.90 (6.99) | 1.18 (10.46) | -1.53 (6.48) | -0.46 (8.49)
  ALT, Day 15: number analyzed (Participants) | 36 | 35 | 39 | 32 | 38
  ALT, Day 15 | 1.03 (15.17) | -0.54 (7.99) | -0.21 (10.54) | -2.69 (6.69) | -1.95 (8.92)
  ALT, Day 22: number analyzed (Participants) | 39 | 37 | 39 | 33 | 38
  ALT, Day 22 | 0.13 (13.64) | 3.05 (13.37) | -0.41 (10.98) | -0.21 (9.78) | -3.71 (11.15)
  ALT, Day 28: number analyzed (Participants) | 39 | 32 | 36 | 30 | 36
  ALT, Day 28 | -2.79 (11.14) | 0.56 (13.18) | -0.47 (13.17) | -2.27 (9.81) | -3.86 (11.10)
  ALT, Day 35: number analyzed (Participants) | 37 | 40 | 39 | 32 | 40
  ALT, Day 35 | -2.49 (11.86) | -0.38 (9.43) | -0.97 (10.85) | -3.06 (9.14) | -3.13 (11.78)
  ALP, Day 8: number analyzed (Participants) | 41 | 41 | 40 | 37 | 41
  ALP, Day 8 | -3.22 (7.60) | -0.63 (9.80) | -1.60 (8.15) | -3.24 (9.00) | 0.63 (9.90)
  ALP, Day 15: number analyzed (Participants) | 38 | 36 | 41 | 36 | 40
  ALP, Day 15 | -1.61 (15.02) | -4.17 (14.55) | -2.05 (12.83) | -5.67 (18.08) | -1.65 (10.35)
  ALP, Day 22: number analyzed (Participants) | 41 | 38 | 41 | 36 | 40
  ALP, Day 22 | -3.17 (10.10) | -0.55 (17.35) | -0.22 (13.95) | -2.08 (19.56) | -2.20 (12.29)
  ALP, Day 28: number analyzed (Participants) | 41 | 35 | 40 | 36 | 39
  ALP, Day 28 | -4.73 (12.20) | -1.34 (19.89) | -3.33 (14.41) | -4.61 (18.06) | -4.05 (15.79)
  ALP, Day 35: number analyzed (Participants) | 39 | 41 | 41 | 35 | 42
  ALP, Day 35 | -5.95 (12.74) | -2.10 (15.76) | -2.71 (13.71) | -6.34 (16.37) | -4.69 (16.79)
  AST, Day 8: number analyzed (Participants) | 39 | 40 | 38 | 34 | 39
  AST, Day 8 | -1.33 (10.28) | -1.25 (6.30) | -0.63 (6.92) | -1.18 (10.44) | 0.46 (4.89)
  AST, Day 15: number analyzed (Participants) | 36 | 35 | 39 | 33 | 38
  AST, Day 15 | -0.97 (13.71) | -0.54 (6.27) | -0.38 (9.60) | -2.85 (11.39) | 0.37 (5.27)
  AST, Day 22: number analyzed (Participants) | 39 | 36 | 39 | 34 | 38
  AST, Day 22 | -1.36 (11.82) | 1.47 (6.43) | -0.95 (11.51) | -0.97 (12.87) | -1.50 (6.33)
  AST, Day 28: number analyzed (Participants) | 39 | 31 | 36 | 30 | 36
  AST, Day 28 | -2.28 (11.28) | -1.39 (6.93) | -0.69 (9.92) | -2.23 (11.76) | -1.44 (4.95)
  AST, Day 35: number analyzed (Participants) | 37 | 40 | 38 | 33 | 40
  AST, Day 35 | -2.14 (11.95) | -1.38 (6.52) | -0.82 (10.05) | -1.88 (12.15) | -1.88 (5.21)
  Creatinine phosphokinase, Day 8: number analyzed (Participants) | 39 | 40 | 39 | 35 | 41
  Creatinine phosphokinase, Day 8 | -4.05 (30.14) | 11.25 (79.26) | -10.95 (84.04) | -3.11 (30.12) | -8.37 (100.00)
  Creatinine phosphokinase, Day 15: number analyzed (Participants) | 36 | 35 | 40 | 34 | 40
  Creatinine phosphokinase, Day 15 | -9.03 (39.62) | 4.46 (33.64) | -10.23 (77.79) | -7.06 (43.44) | -0.05 (101.77)
  Creatinine phosphokinase, Day 22: number analyzed (Participants) | 39 | 37 | 40 | 34 | 40
  Creatinine phosphokinase, Day 22 | 0.28 (33.55) | 27.54 (97.86) | -19.40 (74.31) | 6.47 (33.44) | -9.18 (100.75)
  Creatinine phosphokinase, Day 28: number analyzed (Participants) | 39 | 33 | 36 | 34 | 38
  Creatinine phosphokinase, Day 28 | -3.74 (51.30) | 2.61 (32.25) | -15.03 (84.44) | 12.65 (40.68) | -3.47 (110.21)
  Creatinine phosphokinase, Day 35: number analyzed (Participants) | 37 | 40 | 40 | 33 | 42
  Creatinine phosphokinase, Day 35 | -4.65 (23.19) | 0.38 (31.87) | -12.58 (82.07) | 8.30 (33.05) | -4.33 (104.54)
  LDH, Day 8: number analyzed (Participants) | 37 | 34 | 37 | 30 | 35
  LDH, Day 8 | -9.27 (55.02) | 0.03 (20.69) | 1.51 (20.44) | -5.23 (18.38) | -0.54 (14.93)
  LDH, Day 15: number analyzed (Participants) | 35 | 31 | 38 | 32 | 36
  LDH, Day 15 | -3.31 (52.15) | 0.58 (20.51) | -2.45 (23.63) | -6.09 (29.60) | -2.64 (16.74)
  LDH, Day 22: number analyzed (Participants) | 37 | 30 | 38 | 31 | 36
  LDH, Day 22 | -8.84 (58.19) | -0.33 (21.26) | -2.34 (22.19) | -3.61 (22.03) | -3.42 (16.53)
  LDH, Day 28: number analyzed (Participants) | 37 | 27 | 32 | 27 | 31
  LDH, Day 28 | -11.27 (56.13) | -5.04 (19.71) | -7.44 (18.31) | -6.70 (16.99) | -1.48 (16.83)
  LDH, Day 35: number analyzed (Participants) | 34 | 35 | 37 | 31 | 38
  LDH, Day 35 | -7.47 (60.72) | -1.74 (20.90) | 2.19 (25.99) | -1.65 (23.37) | -3.68 (16.18)

19. Primary Outcome: Change From Baseline in Chemistry Parameter of Bicarbonate, Blood Urea Nitrogen (BUN), Calcium, Chloride, Magnesium, Phosphate, Potassium and Sodium Over Time
Description: Assessment for bicarbonate, BUN, calcium, chloride, magnesium, phosphate, potassium and sodium were performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromole (mmol) per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Micromole (mmol) per liter
  Bicarbonate, Day 8: number analyzed (Participants) | 42 | 41 | 39 | 38 | 41
  Bicarbonate, Day 8 | 0.74 (2.69) | 0.78 (3.01) | 0.62 (2.40) | 0.13 (2.48) | -0.17 (2.64)
  Bicarbonate, Day 15: number analyzed (Participants) | 41 | 36 | 41 | 38 | 39
  Bicarbonate, Day 15 | 0.85 (2.36) | 1.47 (2.68) | 0.41 (2.45) | 0.42 (2.52) | 0.03 (2.86)
  Bicarbonate, Day 22: number analyzed (Participants) | 43 | 38 | 41 | 38 | 40
  Bicarbonate, Day 22 | 0.65 (2.71) | 1.45 (2.69) | 0.90 (2.96) | 0.03 (2.49) | 0.00 (2.60)
  Bicarbonate, Day 28: number analyzed (Participants) | 43 | 35 | 41 | 38 | 40
  Bicarbonate, Day 28 | -0.09 (2.61) | 0.40 (2.66) | -0.37 (2.67) | -0.13 (2.42) | -0.68 (1.97)
  Bicarbonate, Day 35: number analyzed (Participants) | 41 | 41 | 42 | 36 | 42
  Bicarbonate, Day 35 | 0.68 (2.96) | 0.51 (2.61) | 0.60 (2.65) | -0.14 (2.31) | -0.48 (2.75)
  BUN, Day 8: number analyzed (Participants) | 42 | 41 | 41 | 39 | 41
  BUN, Day 8 | -0.09 (1.40) | 0.30 (2.05) | 0.29 (1.39) | 0.15 (1.40) | 0.03 (1.19)
  BUN, Day 15: number analyzed (Participants) | 39 | 36 | 42 | 38 | 40
  BUN, Day 15 | -0.06 (1.43) | 0.16 (2.19) | 0.15 (1.00) | 0.42 (1.33) | 0.36 (1.46)
  BUN, Day 22: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  BUN, Day 22 | -0.03 (1.21) | 0.36 (2.01) | 0.27 (1.16) | 0.01 (1.46) | 0.16 (1.16)
  BUN, Day 28: number analyzed (Participants) | 42 | 35 | 41 | 38 | 40
  BUN, Day 28 | 0.25 (1.39) | 0.91 (2.11) | 0.24 (1.29) | -0.15 (1.49) | 0.09 (1.25)
  BUN, Day 35: number analyzed (Participants) | 40 | 41 | 42 | 37 | 42
  BUN, Day 35 | -0.07 (1.51) | 0.35 (1.78) | 0.22 (1.40) | -0.57 (1.37) | -0.11 (1.40)
  Calcium, Day 8: number analyzed (Participants) | 41 | 41 | 41 | 39 | 41
  Calcium, Day 8 | 0.03 (0.09) | 0.02 (0.12) | 0.03 (0.11) | 0.05 (0.10) | 0.02 (0.09)
  Calcium, Day 15: number analyzed (Participants) | 38 | 36 | 42 | 38 | 40
  Calcium, Day 15 | 0.04 (0.10) | 0.00 (0.15) | 0.01 (0.10) | 0.05 (0.12) | -0.01 (0.10)
  Calcium, Day 22: number analyzed (Participants) | 41 | 38 | 42 | 38 | 40
  Calcium, Day 22 | 0.02 (0.08) | 0.01 (0.13) | 0.01 (0.10) | 0.05 (0.08) | -0.00 (0.09)
  Calcium, Day 28: number analyzed (Participants) | 41 | 35 | 41 | 38 | 40
  Calcium, Day 28 | 0.00 (0.11) | -0.02 (0.15) | -0.03 (0.12) | 0.02 (0.11) | -0.04 (0.10)
  Calcium, Day 35: number analyzed (Participants) | 39 | 41 | 42 | 37 | 42
  Calcium, Day 35 | 0.02 (0.11) | -0.01 (0.11) | -0.00 (0.09) | 0.02 (0.08) | -0.02 (0.11)
  Chloride, Day 8: number analyzed (Participants) | 42 | 42 | 41 | 41 | 41
  Chloride, Day 8 | 0.45 (2.44) | -0.14 (3.07) | 0.46 (2.96) | 0.12 (2.82) | -0.80 (2.72)
  Chloride, Day 15: number analyzed (Participants) | 41 | 40 | 42 | 41 | 41
  Chloride, Day 15 | 0.24 (3.01) | 0.00 (3.16) | 0.29 (2.63) | 0.90 (2.50) | -0.71 (3.39)
  Chloride, Day 22: number analyzed (Participants) | 42 | 39 | 42 | 40 | 40
  Chloride, Day 22 | 0.57 (2.61) | -0.26 (3.27) | 0.45 (2.98) | 1.10 (3.11) | -0.65 (3.00)
  Chloride, Day 28: number analyzed (Participants) | 42 | 36 | 41 | 40 | 40
  Chloride, Day 28 | -0.17 (2.78) | 0.17 (3.30) | 0.54 (3.06) | 0.43 (3.27) | 0.00 (3.45)
  Chloride, Day 35: number analyzed (Participants) | 41 | 42 | 42 | 40 | 42
  Chloride, Day 35 | 0.49 (3.00) | 0.98 (2.88) | 1.40 (3.00) | 1.38 (3.13) | 0.95 (3.09)
  Magnesium, Day 8: number analyzed (Participants) | 41 | 41 | 40 | 37 | 41
  Magnesium, Day 8 | 0.01 (0.07) | 0.00 (0.06) | -0.02 (0.06) | -0.01 (0.06) | 0.01 (0.06)
  Magnesium, Day 15: number analyzed (Participants) | 39 | 37 | 41 | 36 | 40
  Magnesium, Day 15 | 0.01 (0.06) | -0.01 (0.07) | -0.01 (0.06) | -0.01 (0.06) | -0.00 (0.04)
  Magnesium, Day 22: number analyzed (Participants) | 41 | 38 | 41 | 36 | 40
  Magnesium, Day 22 | 0.01 (0.08) | 0.00 (0.07) | -0.01 (0.06) | 0.00 (0.06) | -0.00 (0.08)
  Magnesium, Day 28: number analyzed (Participants) | 41 | 35 | 40 | 36 | 39
  Magnesium, Day 28 | 0.00 (0.06) | -0.01 (0.06) | -0.02 (0.06) | 0.01 (0.06) | -0.01 (0.05)
  Magnesium, Day 35: number analyzed (Participants) | 40 | 41 | 41 | 35 | 42
  Magnesium, Day 35 | -0.01 (0.06) | -0.02 (0.08) | -0.01 (0.06) | -0.00 (0.08) | -0.00 (0.07)
  Phosphate, Day 8: number analyzed (Participants) | 42 | 41 | 40 | 38 | 41
  Phosphate, Day 8 | -0.02 (0.21) | -0.02 (0.19) | -0.00 (0.18) | -0.03 (0.20) | 0.03 (0.13)
  Phosphate, Day 15: number analyzed (Participants) | 39 | 36 | 41 | 37 | 40
  Phosphate, Day 15 | 0.04 (0.21) | -0.01 (0.16) | -0.01 (0.15) | -0.04 (0.20) | -0.01 (0.17)
  Phosphate, Day 22: number analyzed (Participants) | 42 | 38 | 41 | 37 | 40
  Phosphate, Day 22 | 0.01 (0.21) | 0.04 (0.19) | -0.01 (0.16) | -0.03 (0.22) | -0.00 (0.18)
  Phosphate, Day 28: number analyzed (Participants) | 42 | 35 | 40 | 37 | 39
  Phosphate, Day 28 | -0.00 (0.20) | -0.00 (0.19) | 0.02 (0.18) | -0.03 (0.22) | -0.00 (0.16)
  Phosphate, Day 35: number analyzed (Participants) | 40 | 41 | 41 | 36 | 42
  Phosphate, Day 35 | -0.00 (0.20) | -0.04 (0.18) | -0.01 (0.14) | -0.02 (0.23) | 0.04 (0.21)
  Potassium, Day 8: number analyzed (Participants) | 39 | 41 | 39 | 37 | 41
  Potassium, Day 8 | 0.29 (0.48) | 0.11 (0.38) | 0.27 (0.45) | 0.24 (0.47) | 0.19 (0.42)
  Potassium, Day 15: number analyzed (Participants) | 38 | 39 | 40 | 37 | 41
  Potassium, Day 15 | 0.23 (0.46) | 0.16 (0.35) | 0.25 (0.41) | 0.34 (0.47) | 0.13 (0.35)
  Potassium, Day 22: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Potassium, Day 22 | 0.19 (0.53) | 0.13 (0.40) | 0.28 (0.41) | 0.31 (0.51) | 0.14 (0.40)
  Potassium, Day 28: number analyzed (Participants) | 39 | 33 | 36 | 36 | 38
  Potassium, Day 28 | 0.00 (0.43) | -0.02 (0.52) | 0.07 (0.37) | 0.03 (0.48) | -0.20 (0.31)
  Potassium, Day 35: number analyzed (Participants) | 38 | 41 | 40 | 36 | 42
  Potassium, Day 35 | 0.25 (0.59) | 0.07 (0.45) | 0.23 (0.35) | 0.20 (0.44) | 0.10 (0.42)
  Sodium, Day 8: number analyzed (Participants) | 42 | 42 | 41 | 41 | 41
  Sodium, Day 8 | 0.05 (2.48) | -0.33 (2.72) | 0.29 (2.62) | 0.05 (2.93) | -0.41 (2.74)
  Sodium, Day 15: number analyzed (Participants) | 41 | 40 | 42 | 41 | 41
  Sodium, Day 15 | 0.10 (3.08) | -0.53 (2.69) | -0.31 (2.57) | 0.80 (2.90) | -0.59 (3.19)
  Sodium, Day 22: number analyzed (Participants) | 42 | 39 | 42 | 40 | 40
  Sodium, Day 22 | 0.31 (2.42) | -0.46 (2.34) | 0.29 (2.80) | 1.03 (3.06) | -0.63 (2.83)
  Sodium, Day 28: number analyzed (Participants) | 42 | 36 | 41 | 40 | 40
  Sodium, Day 28 | 0.07 (2.87) | -0.11 (3.35) | -0.15 (2.82) | 0.73 (2.67) | -0.40 (3.09)
  Sodium, Day 35: number analyzed (Participants) | 41 | 42 | 42 | 40 | 42
  Sodium, Day 35 | 0.71 (2.94) | 0.07 (2.78) | 0.57 (3.01) | 1.10 (2.33) | 0.24 (2.41)

20. Primary Outcome: Change From Baseline in Chemistry Parameter of Direct Bilirubin, Indirect Bilirubin, Serum Creatinine, Total Bilirubin and Uric Acid Over Time
Description: Assessment for direct bilirubin, indirect bilirubin, serum creatinine, total bilirubin and uric acid were performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromole per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Micromole per liter
  Direct bilirubin, Day 8: number analyzed (Participants) | 37 | 35 | 37 | 32 | 37
  Direct bilirubin, Day 8 | -0.05 (0.88) | 0.26 (0.78) | 0.27 (0.65) | 0.13 (0.55) | 0.30 (0.88)
  Direct bilirubin, Day 15: number analyzed (Participants) | 35 | 31 | 39 | 31 | 37
  Direct bilirubin, Day 15 | 0.11 (0.68) | 0.19 (0.60) | 0.13 (0.52) | -0.06 (0.44) | 0.43 (0.90)
  Direct bilirubin, Day 22: number analyzed (Participants) | 37 | 31 | 39 | 32 | 38
  Direct bilirubin, Day 22 | 0.19 (0.70) | 0.10 (0.70) | 0.08 (0.35) | 0.03 (0.74) | 0.21 (0.58)
  Direct bilirubin, Day 28: number analyzed (Participants) | 38 | 28 | 32 | 28 | 35
  Direct bilirubin, Day 28 | -0.08 (0.59) | 0.07 (0.38) | 0.19 (0.74) | -0.11 (0.50) | 0.26 (0.85)
  Direct bilirubin, Day 35: number analyzed (Participants) | 34 | 34 | 38 | 32 | 37
  Direct bilirubin, Day 35 | -0.06 (0.92) | -0.06 (0.60) | -0.05 (0.32) | -0.25 (0.67) | 0.00 (0.53)
  Indirect bilirubin, Day 8: number analyzed (Participants) | 37 | 35 | 37 | 32 | 37
  Indirect bilirubin, Day 8 | -0.30 (3.02) | 1.06 (3.31) | 1.49 (3.52) | 0.91 (3.32) | 1.22 (4.36)
  Indirect bilirubin, Day 15: number analyzed (Participants) | 35 | 31 | 39 | 31 | 37
  Indirect bilirubin, Day 15 | 0.31 (2.47) | 0.71 (4.03) | 0.56 (2.55) | 0.52 (3.37) | 1.22 (2.90)
  Indirect bilirubin, Day 22: number analyzed (Participants) | 37 | 31 | 39 | 32 | 38
  Indirect bilirubin, Day 22 | 0.70 (3.44) | 0.61 (3.04) | 0.62 (3.27) | 1.09 (3.37) | 0.39 (2.69)
  Indirect bilirubin, Day 28: number analyzed (Participants) | 38 | 28 | 32 | 28 | 35
  Indirect bilirubin, Day 28 | -0.58 (3.59) | 0.04 (3.21) | 0.38 (2.69) | -0.36 (2.68) | -0.37 (3.53)
  Indirect bilirubin, Day 35: number analyzed (Participants) | 34 | 34 | 38 | 32 | 37
  Indirect bilirubin, Day 35 | -0.38 (3.37) | -0.38 (3.56) | -0.08 (2.95) | -1.63 (3.90) | -1.24 (2.78)
  Serum creatinine, Day 8: number analyzed (Participants) | 42 | 41 | 41 | 39 | 41
  Serum creatinine, Day 8 | 0.31 (6.78) | 1.68 (8.98) | 4.27 (8.20) | 5.26 (9.20) | 7.15 (10.89)
  Serum creatinine, Day 15: number analyzed (Participants) | 39 | 36 | 42 | 38 | 40
  Serum creatinine, Day 15 | -1.05 (6.80) | 1.00 (8.91) | 2.21 (6.97) | 2.45 (8.30) | 5.83 (10.15)
  Serum creatinine, Day 22: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Serum creatinine, Day 22 | -0.74 (6.97) | 1.13 (10.01) | 2.57 (7.17) | 2.61 (9.49) | 5.50 (8.23)
  Serum creatinine, Day 28: number analyzed (Participants) | 42 | 35 | 41 | 38 | 40
  Serum creatinine, Day 28 | -1.12 (7.38) | 1.09 (9.24) | 1.85 (9.47) | 1.03 (6.89) | 2.78 (9.16)
  Serum creatinine, Day 35: number analyzed (Participants) | 40 | 41 | 42 | 37 | 42
  Serum creatinine, Day 35 | -0.75 (7.50) | 0.07 (9.91) | 0.93 (6.87) | -1.46 (6.89) | 0.40 (8.00)
  Total bilirubin, Day 8: number analyzed (Participants) | 41 | 41 | 39 | 38 | 39
  Total bilirubin, Day 8 | -0.49 (3.72) | 1.24 (3.73) | 1.77 (4.13) | 1.39 (3.78) | 2.08 (6.16)
  Total bilirubin, Day 15: number analyzed (Participants) | 39 | 36 | 41 | 37 | 39
  Total bilirubin, Day 15 | 0.44 (3.16) | 1.25 (4.16) | 0.73 (2.95) | 1.68 (4.87) | 1.95 (4.42)
  Total bilirubin, Day 22: number analyzed (Participants) | 41 | 38 | 41 | 38 | 39
  Total bilirubin, Day 22 | 0.98 (3.75) | 1.05 (3.38) | 0.83 (3.41) | 1.76 (3.97) | 1.21 (4.57)
  Total bilirubin, Day 28: number analyzed (Participants) | 42 | 35 | 39 | 37 | 39
  Total bilirubin, Day 28 | -0.64 (4.17) | 0.17 (3.46) | 0.90 (3.39) | 0.30 (4.22) | -0.03 (5.22)
  Total bilirubin, Day 35: number analyzed (Participants) | 39 | 39 | 41 | 37 | 38
  Total bilirubin, Day 35 | -0.62 (4.24) | -0.33 (3.72) | -0.32 (3.39) | -1.81 (5.34) | -1.39 (3.28)
  Uric acid, Day 8: number analyzed (Participants) | 42 | 41 | 40 | 39 | 41
  Uric acid, Day 8 | 1.38 (38.94) | -8.66 (55.20) | -22.90 (48.36) | -20.95 (61.72) | -26.20 (66.02)
  Uric acid, Day 15: number analyzed (Participants) | 39 | 36 | 41 | 38 | 40
  Uric acid, Day 15 | -5.95 (59.07) | -13.19 (54.16) | -20.29 (39.59) | -11.13 (74.79) | -7.70 (63.59)
  Uric acid, Day 22: number analyzed (Participants) | 42 | 38 | 41 | 38 | 40
  Uric acid, Day 22 | -1.40 (46.23) | -3.55 (53.46) | -21.63 (52.20) | -13.61 (57.87) | -13.88 (70.17)
  Uric acid, Day 28: number analyzed (Participants) | 42 | 35 | 40 | 38 | 40
  Uric acid, Day 28 | 5.69 (50.16) | 6.20 (74.17) | -10.73 (41.62) | -6.00 (61.23) | -18.05 (82.41)
  Uric acid, Day 35: number analyzed (Participants) | 40 | 41 | 41 | 37 | 42
  Uric acid, Day 35 | 2.30 (55.55) | -8.63 (57.75) | -4.51 (56.60) | 12.03 (59.59) | -2.45 (57.67)

21. Primary Outcome: Change From Baseline in Chemistry Parameter of Lipid Profile Over Time
Description: Assessment for lipid profile was performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. The parameters included high density lipoprotein (HDL), low density lipoprotein (LDL), total cholesterol and triglycerides. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
mmol per liter
  HDL, Day 8: number analyzed (Participants) | 42 | 41 | 41 | 39 | 41
  HDL, Day 8 | -0.02 (0.14) | 0.01 (0.19) | 0.02 (0.19) | 0.05 (0.18) | -0.03 (0.17)
  HDL, Day 15: number analyzed (Participants) | 39 | 36 | 42 | 38 | 40
  HDL, Day 15 | -0.02 (0.21) | 0.01 (0.17) | -0.01 (0.20) | 0.08 (0.21) | -0.03 (0.16)
  HDL, Day 22: number analyzed (Participants) | 42 | 38 | 41 | 38 | 40
  HDL, Day 22 | -0.03 (0.21) | 0.02 (0.23) | 0.02 (0.19) | 0.05 (0.14) | -0.04 (0.18)
  HDL, Day 28: number analyzed (Participants) | 42 | 35 | 41 | 38 | 40
  HDL, Day 28 | -0.04 (0.24) | -0.02 (0.20) | -0.04 (0.20) | 0.01 (0.18) | -0.05 (0.20)
  HDL, Day 35: number analyzed (Participants) | 40 | 41 | 42 | 37 | 42
  HDL, Day 35 | -0.03 (0.22) | 0.00 (0.17) | -0.01 (0.22) | 0.05 (0.15) | -0.01 (0.18)
  LDL, Day 8: number analyzed (Participants) | 40 | 41 | 41 | 38 | 41
  LDL, Day 8 | -0.10 (0.57) | -0.27 (0.76) | -0.16 (0.57) | -0.19 (0.45) | -0.20 (0.51)
  LDL, Day 15: number analyzed (Participants) | 38 | 36 | 42 | 37 | 40
  LDL, Day 15 | -0.07 (0.53) | -0.26 (0.83) | -0.23 (0.76) | -0.22 (0.61) | -0.26 (0.59)
  LDL, Day 22: number analyzed (Participants) | 41 | 38 | 41 | 37 | 40
  LDL, Day 22 | -0.02 (0.68) | -0.34 (0.67) | -0.14 (0.88) | -0.23 (0.52) | -0.17 (0.74)
  LDL, Day 28: number analyzed (Participants) | 41 | 35 | 41 | 37 | 39
  LDL, Day 28 | -0.07 (0.69) | -0.17 (0.77) | -0.29 (0.75) | -0.28 (0.59) | -0.22 (0.86)
  LDL, Day 35: number analyzed (Participants) | 39 | 40 | 42 | 36 | 42
  LDL, Day 35 | -0.08 (0.71) | -0.30 (0.83) | -0.14 (0.77) | -0.15 (0.50) | -0.07 (0.86)
  Total cholesterol, Day 8: number analyzed (Participants) | 41 | 41 | 41 | 39 | 41
  Total cholesterol, Day 8 | -0.16 (0.62) | -0.33 (0.89) | -0.27 (0.72) | -0.38 (0.50) | -0.27 (0.59)
  Total cholesterol, Day 15: number analyzed (Participants) | 38 | 36 | 42 | 38 | 40
  Total cholesterol, Day 15 | -0.09 (0.71) | -0.38 (0.97) | -0.27 (0.98) | -0.35 (0.82) | -0.27 (0.72)
  Total cholesterol, Day 22: number analyzed (Participants) | 41 | 38 | 41 | 38 | 40
  Total cholesterol, Day 22 | -0.09 (0.92) | -0.46 (0.81) | -0.16 (1.06) | -0.49 (0.81) | -0.20 (0.88)
  Total cholesterol, Day 28: number analyzed (Participants) | 41 | 35 | 41 | 38 | 40
  Total cholesterol, Day 28 | -0.15 (0.97) | -0.23 (0.93) | -0.25 (0.89) | -0.55 (0.81) | -0.23 (0.92)
  Total cholesterol, Day 35: number analyzed (Participants) | 39 | 41 | 42 | 37 | 42
  Total cholesterol, Day 35 | -0.11 (0.98) | -0.47 (0.88) | -0.22 (1.07) | -0.41 (0.93) | -0.11 (1.04)
  Triglycerides, Day 8: number analyzed (Participants) | 42 | 41 | 41 | 38 | 41
  Triglycerides, Day 8 | -0.15 (0.93) | -0.14 (1.12) | -0.22 (0.76) | -0.66 (1.33) | -0.13 (0.63)
  Triglycerides, Day 15: number analyzed (Participants) | 39 | 36 | 42 | 37 | 40
  Triglycerides, Day 15 | 0.04 (1.05) | -0.34 (1.36) | 0.02 (1.23) | -0.50 (0.97) | 0.07 (1.02)
  Triglycerides, Day 22: number analyzed (Participants) | 42 | 38 | 41 | 37 | 40
  Triglycerides, Day 22 | -0.08 (1.03) | -0.36 (1.30) | -0.02 (0.97) | -0.83 (1.89) | 0.08 (1.32)
  Triglycerides, Day 28: number analyzed (Participants) | 42 | 35 | 41 | 37 | 39
  Triglycerides, Day 28 | -0.08 (1.06) | -0.09 (1.60) | 0.22 (0.95) | -0.75 (1.91) | 0.03 (1.51)
  Triglycerides, Day 35: number analyzed (Participants) | 40 | 41 | 42 | 36 | 42
  Triglycerides, Day 35 | -0.02 (0.83) | -0.30 (0.81) | -0.32 (3.03) | -0.90 (2.29) | -0.19 (0.88)

22. Primary Outcome: Change From Baseline in Chemistry Parameter of Albumin and Total Protein Over Time
Description: Assessment for albumin and total protein were performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Gram per liter
  Albumin, Day 8: number analyzed (Participants) | 42 | 41 | 41 | 39 | 41
  Albumin, Day 8 | 0.29 (2.03) | 0.80 (2.40) | 0.78 (2.72) | 0.64 (2.05) | 1.02 (1.93)
  Albumin, Day 15: number analyzed (Participants) | 40 | 37 | 42 | 38 | 40
  Albumin, Day 15 | 0.80 (2.44) | 1.05 (2.39) | 0.29 (2.39) | 0.13 (2.24) | 0.53 (2.06)
  Albumin, Day 22: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Albumin, Day 22 | 0.67 (1.91) | 0.82 (2.46) | 0.10 (2.34) | 0.55 (2.37) | 0.40 (2.02)
  Albumin, Day 28: number analyzed (Participants) | 42 | 35 | 41 | 38 | 40
  Albumin, Day 28 | 0.45 (2.15) | 0.00 (2.45) | -0.63 (2.79) | -0.32 (2.24) | -0.53 (2.40)
  Albumin, Day 35: number analyzed (Participants) | 41 | 41 | 42 | 37 | 42
  Albumin, Day 35 | -0.02 (2.59) | -0.07 (2.08) | -0.17 (2.56) | -0.16 (2.48) | -0.21 (2.31)
  Total protein, Day 8: number analyzed (Participants) | 42 | 41 | 40 | 39 | 41
  Total protein, Day 8 | -0.24 (3.33) | 1.24 (4.39) | 0.23 (4.29) | 0.21 (3.15) | 1.24 (4.16)
  Total protein, Day 15: number analyzed (Participants) | 39 | 36 | 41 | 38 | 40
  Total protein, Day 15 | 0.44 (4.43) | 0.67 (4.68) | 0.63 (4.92) | -1.24 (4.28) | -0.03 (4.38)
  Total protein, Day 22: number analyzed (Participants) | 42 | 38 | 41 | 38 | 40
  Total protein, Day 22 | 0.48 (3.21) | 1.29 (5.54) | 0.49 (4.90) | 0.18 (3.81) | -0.03 (3.88)
  Total protein, Day 28: number analyzed (Participants) | 42 | 35 | 40 | 38 | 39
  Total protein, Day 28 | 0.21 (3.76) | 0.06 (5.17) | -1.10 (5.45) | -0.63 (3.76) | -1.49 (4.48)
  Total protein, Day 35: number analyzed (Participants) | 40 | 41 | 41 | 37 | 42
  Total protein, Day 35 | -0.05 (4.03) | -0.61 (3.94) | -0.07 (4.66) | -0.95 (4.16) | -1.57 (4.80)

23. Primary Outcome: Change From Baseline in Urinalysis Parameter of Specific Gravity Over Time
Description: Urinary specific gravity is a measure of the concentration of solutes in urine. It measures the ratio of urine density compared with water density and provides information on the kidney's ability to concentrate urine. The assessments were performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Ratio
  Day 8: number analyzed (Participants) | 42 | 41 | 41 | 38 | 38
  Day 8 | -0.00 (0.01) | -0.00 (0.01) | 0.00 (0.01) | -0.00 (0.01) | -0.00 (0.01)
  Day 15: number analyzed (Participants) | 41 | 36 | 41 | 37 | 39
  Day 15 | -0.00 (0.01) | -0.00 (0.00) | -0.00 (0.01) | -0.00 (0.01) | 0.00 (0.01)
  Day 22: number analyzed (Participants) | 43 | 37 | 42 | 38 | 39
  Day 22 | -0.00 (0.01) | -0.00 (0.01) | 0.00 (0.01) | -0.00 (0.01) | 0.00 (0.01)
  Day 28: number analyzed (Participants) | 43 | 35 | 42 | 37 | 39
  Day 28 | 0.00 (0.01) | -0.00 (0.01) | 0.00 (0.01) | -0.00 (0.01) | 0.00 (0.01)
  Day 35: number analyzed (Participants) | 39 | 39 | 43 | 37 | 39
  Day 35 | -0.00 (0.01) | -0.00 (0.01) | 0.00 (0.01) | -0.00 (0.01) | -0.00 (0.01)

24. Primary Outcome: Change From Baseline in Urinalysis Parameter of pH Over Time
Description: Urinalysis parameter included urine pH. pH was calculated on a scale of 0 to 14, such that, the lower the number, more acidic the urine and higher the number, more alkaline the urine with 7 being neutral. The assessment was performed on Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: Safety Analysis Set Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 43 | 44 | 42 | 43
Points on scale
  Day 8: number analyzed (Participants) | 43 | 41 | 41 | 39 | 40
  Day 8 | 0.05 (0.34) | -0.05 (0.38) | -0.02 (0.35) | 0.00 (0.43) | 0.10 (0.51)
  Day 15: number analyzed (Participants) | 41 | 36 | 41 | 38 | 40
  Day 15 | 0.05 (0.35) | -0.04 (0.45) | -0.05 (0.57) | 0.11 (0.47) | 0.08 (0.62)
  Day 22: number analyzed (Participants) | 43 | 37 | 42 | 38 | 40
  Day 22 | 0.14 (0.41) | -0.03 (0.50) | 0.01 (0.55) | 0.05 (0.40) | -0.03 (0.48)
  Day 28: number analyzed (Participants) | 43 | 35 | 42 | 38 | 40
  Day 28 | 0.28 (0.66) | -0.09 (0.43) | 0.00 (0.59) | 0.03 (0.37) | 0.04 (0.63)
  Day 35: number analyzed (Participants) | 39 | 41 | 43 | 37 | 42
  Day 35 | 0.06 (0.48) | -0.15 (0.37) | -0.12 (0.55) | 0.01 (0.38) | 0.07 (0.52)

25. Primary Outcome: Area Under Plasma Concentration Curve From Time 0 to Last Measurable Time Point (AUC 0-t), From Time 0 to Infinity (AUC 0-infinity) and From Time 0 to Trough Concentration (AUC 0-τ) of SRT2104 on Day 1 and Day 28
Description: The pre-dose blood samples were collected within one hour prior to study medication administration. The post-dose blood samples were collected within 2 minutes of the scheduled time. AUC values reported in the analysis of AUC 0-infinity of Day 28 versus Day 1 included AUC 0-infinity on Day 1 and AUC 0-τ on Day 28. Participants fasted for at least 10 hour overnight on Day 1, 2 and 29. The AUC 0-t was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. AUC0-infinity was estimated by linear trapezoidal rule and was sum of the AUC0-t and extrapolated to infinity by dividing the estimated last measurable plasma concentration by elimination rate constant lambda z. Where lambda z is the terminal phase rate constant estimated by linear regression analysis of the log10 transformed concentration-time data after each single dose. The AUC0-infinity was the sum of the estimated and extrapolated parts.
Time Frame: Day 1 (pre-dose, 15 and 30 minutes, 1, 2, 3, 4, 8 and 12 hour post-dose), Day 2 (24 hour post-Day 1 dose), Day 8, 15 and 22 (pre-dose), Day 28 (pre-dose, and 15 and 30 minutes, 1, 2, 3, 4, 8 and 12 hour post-dose) and Day 29 (24 hour post-Day 28)
Population: Pharmacokinetic (PK) Population defined as all participants who received SRT2104, had sufficient blood samples taken to obtain a plasma concentration time profile and who did not violate the protocol in such a way that it could influence the statistical analysis. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram (ng)*hour/milliliter (mL)
Arm/Group | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 44 | 42 | 43
Nanogram (ng)*hour/milliliter (mL)
  Day 1, AUC 0-t: number analyzed (Participants) | 39 | 42 | 40 | 40
  Day 1, AUC 0-t | 1045.8420 (978.3355) | 2153.0075 (1835.6039) | 2375.3150 (2285.7123) | 2859.5465 (2916.4783)
  Day 28, AUC 0-t: number analyzed (Participants) | 37 | 42 | 40 | 40
  Day 28, AUC 0-t | 1549.6139 (1450.1354) | 2731.6308 (2337.0839) | 3109.8747 (2948.2780) | 4380.2204 (4476.9484)
  Day 1, AUC 0-infinity: number analyzed (Participants) | 28 | 36 | 30 | 27
  Day 1, AUC 0-infinity | 1564.4905 (1119.3480) | 2797.6930 (2287.3141) | 3080.6902 (2532.8224) | 3837.1384 (4078.6970)
  Day 28, AUC 0-infinity: number analyzed (Participants) | 28 | 34 | 27 | 24
  Day 28, AUC 0-infinity | 2289.6858 (1876.6537) | 4634.3397 (5387.2429) | 4960.3422 (3914.0260) | 8159.4534 (7592.2760)
  Day 28, AUC 0-τ: number analyzed (Participants) | 35 | 42 | 39 | 37
  Day 28, AUC 0-τ | 1620.5989 (1431.4150) | 2731.6231 (2337.0919) | 3212.6640 (2924.1860) | 4584.5679 (4502.8752)
Statistical Analysis 1: Comparison: SRT2104 0.25 g/Day; Day 28 versus Day 1 for AUC 0-t of SRT2104 0.25 g/day; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANOVA; Results obtained from a mixed model ANOVA on log10-transformed data with fixed effect of study day and a random effect of participant; Ratio = 168.40, 90% CI 2-sided [123.87 to 228.94] — The difference in least squares means and corresponding confidence interval (CI) were back-transformed to form ratio of geometric least squares means (Day 28/ Day 1) and CI
Statistical Analysis 2: Comparison: SRT2104 0.25 g/Day; Day 28 versus Day 1 for AUC 0-infinity of SRT2104 0.25 g/day; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANOVA; [statistical method as in outcome 25, analysis 1]; Ratio = 110.88, 90% CI 2-sided [88.18 to 139.43] — The difference in least squares means and corresponding CI were back-transformed to form ratio of geometric least squares means (Day 28/ Day 1) and CI. AUC values included in the analysis were AUC 0-infinity on Day 1 and AUC 0-τ on Day 28
Statistical Analysis 3: Comparison: SRT2104 0.5 g/Day; Day 28 versus Day 1 for AUC 0-t of SRT2104 0.5 g/day; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANOVA; [statistical method as in outcome 25, analysis 1]; Ratio = 133.11, 90% CI 2-sided [100.55 to 176.21] — The difference in least squares means and corresponding CI were back-transformed to form ratio of geometric least squares means (Day 28/ Day 1) and CI
Statistical Analysis 4: Comparison: SRT2104 0.5 g/Day; Day 28 versus Day 1 for AUC 0-infinity of SRT2104 0.5 g/day; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANOVA; [statistical method as in outcome 25, analysis 1]; Other = 94.30, 90% CI 2-sided [70.31 to 126.48] — The difference in least squares means and corresponding CI were back-transformed to form ratio of geometric least squares means (Day 28/ Day 1) and CI. The AUC values included in the analysis were AUC 0-infinity on Day 1 and AUC 0-τ on Day 28
Statistical Analysis 5: Comparison: SRT2104 1.0 g/Day; Day 28 versus Day 1 for AUC 0-t of SRT2104 1.0 g/day; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANOVA; [statistical method as in outcome 25, analysis 1]; Ratio = 141.63, 90% CI 2-sided [111.20 to 180.39] — [estimate comment as in outcome 25, analysis 3]
Statistical Analysis 6: Comparison: SRT2104 1.0 g/Day; Day 28 versus Day 1for AUC 0-infinity of SRT2104 1.0 g/day; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANOVA; [statistical method as in outcome 25, analysis 1]; Ratio = 114.46, 90% CI 2-sided [85.56 to 153.11] — [estimate comment as in outcome 25, analysis 4]
Statistical Analysis 7: Comparison: SRT2104 2.0 g/Day; Day 28 versus Day 1 for AUC 0-t of SRT2104 2.0 g/day; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANOVA; [statistical method as in outcome 25, analysis 1]; Ratio = 167.09, 90% CI 2-sided [120.73 to 231.25] — [estimate comment as in outcome 25, analysis 3]
Statistical Analysis 8: Comparison: SRT2104 2.0 g/Day; Day 28 versus Day 1 for AUC 0-infinity of SRT2104 2.0 g/day; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANOVA; [statistical method as in outcome 25, analysis 1]; Ratio = 117.73, 90% CI 2-sided [85.14 to 162.79] — [estimate comment as in outcome 25, analysis 4]

26. Primary Outcome: Observed Maximum Plasma Concentration (Cmax) of SRT2104 at Day 1 and Day 28
Description: Blood samples were collected on Day 1 (pre-dose, 15 minutes, 30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 8 hour and 12 hour post-dose), Day 2 (24 hour post-Day 1 dose), Day 8 (pre-dose), Day 15 (pre-dose), Day 22 (pre-dose), Day 28 (pre-dose, and 15 minutes, 30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 8 hour and 12 hour post-dose) and Day 29 (24 hour post-Day 28 dose). The pre-dose sample was collected within one hour prior to study medication administration. On Day 1, Day 2 and Day 29, participants fasted for at least 10 hour overnight. The post-dose sample was collected within 2 minutes of the scheduled time. The first occurrence of the Cmax was determined directly from the raw concentration-time data.
Time Frame: Day 1 (pre-dose, 15 and 30 minutes, 1, 2, 3, 4, 8 and 12 hour post-dose), Day 2 (24 hour post-Day 1 dose), Day 8, 15 and 22 (pre-dose), Day 28 (pre-dose, and 15 and 30 minutes, 1, 2, 3, 4, 8 and 12 hour post-dose) and Day 29 (24 hour post-Day 28 dose)
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 44 | 42 | 43
ng/mL
  Day 1: number analyzed (Participants) | 39 | 42 | 40 | 40
  Day 1 | 178.729 (179.982) | 366.694 (322.951) | 336.562 (298.042) | 417.832 (470.048)
  Day 28: number analyzed (Participants) | 38 | 42 | 40 | 40
  Day 28 | 185.418 (162.500) | 329.973 (266.174) | 375.395 (333.188) | 433.650 (461.441)
Statistical Analysis 1: Comparison: SRT2104 0.25 g/Day; Day 28 versus Day 1 for Cmax of SRT2104 0.25 g/day; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANOVA; [statistical method as in outcome 25, analysis 1]; Ratio = 122.22, 90% CI 2-sided [86.94 to 171.80] — [estimate comment as in outcome 25, analysis 3]
Statistical Analysis 2: Comparison: SRT2104 0.5 g/Day; Day 28 versus Day 1 for Cmax of SRT2104 0.5 g/day; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANOVA; [statistical method as in outcome 25, analysis 1]; Ratio = 94.45, 90% CI 2-sided [69.07 to 129.16] — [estimate comment as in outcome 25, analysis 3]
Statistical Analysis 3: Comparison: SRT2104 1.0 g/Day; Day 28 versus Day 1 for Cmax of SRT2104 1.0 g/day; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANOVA; [statistical method as in outcome 25, analysis 1]; Ratio = 114.79, 90% CI 2-sided [91.54 to 143.95] — [estimate comment as in outcome 25, analysis 3]
Statistical Analysis 4: Comparison: SRT2104 2.0 g/Day; Day 28 versus Day 1 for Cmax of SRT2104 2.0 g/day; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANOVA; [statistical method as in outcome 25, analysis 1]; Ratio = 120.30, 90% CI 2-sided [88.66 to 163.23] — [estimate comment as in outcome 25, analysis 3]

27. Primary Outcome: Time to Cmax (Tmax) at Day 1 and Day 28
Description: Blood samples were collected on Day 1 (pre-dose, 15 minutes, 30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 8 hour and 12 hour post-dose), Day 2 (24 hour post-Day 1 dose), Day 8 (pre-dose), Day 15 (pre-dose), Day 22 (pre-dose), Day 28 (pre-dose, and 15 minutes, 30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 8 hour and 12 hour post-dose) and Day 29 (24 hour post-Day 28 dose). The pre-dose sample was collected within one hour prior to study medication administration. The post-dose sample was collected within 2 minutes of the scheduled time. The time at which Cmax was observed was determined directly from the raw concentration-time data.
Time Frame: as for outcome 26
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: hour
Arm/Group | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 44 | 42 | 43
hour
  Day 1: number analyzed (Participants) | 35 | 42 | 40 | 39
  Day 1 | 3.000 [2.000 to 8.000] | 3.000 [1.000 to 24.000] | 3.000 [2.000 to 8.000] | 4.000 [0.250 to 12.000]
  Day 28: number analyzed (Participants) | 36 | 42 | 39 | 38
  Day 28 | 3.000 [0.000 to 24.000] | 3.000 [0.000 to 12.000] | 3.000 [0.000 to 24.000] | 3.000 [0.000 to 12.000]

28. Primary Outcome: Terminal Elimination Half Life (T1/2) of SRT2104 at Day 1 and Day 28
Description: Blood samples were collected on Day 1 (pre-dose, 15 minutes, 30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 8 hour and 12 hour post-dose), Day 2 (24 hour post-Day 1 dose), Day 8 (pre-dose), Day 15 (pre-dose), Day 22 (pre-dose), Day 28 (pre-dose, and 15 minutes, 30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 8 hour and 12 hour post-dose) and Day 29 (24 hour post-Day 28 dose). The pre-dose sample was collected within one hour prior to study medication administration. The post-dose sample was collected within 2 minutes of the scheduled time. On Day 1 Day 2 and Day 29, participants fasted for at least 10 hour overnight. The t1/2 was obtained as the ratio of ln2/λz, where λz is the terminal phase rate constant estimated by linear regression analysis of the concentration-time data.
Time Frame: as for outcome 26
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: hour
Arm/Group | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 44 | 42 | 43
hour
  Day 1: number analyzed (Participants) | 28 | 36 | 30 | 27
  Day 1 | 13.4184 [4.0113 to 33.0069] | 12.1669 [6.1089 to 40.6904] | 13.3434 [6.4721 to 54.7509] | 9.7846 [3.8100 to 24.2013]
  Day 28: number analyzed (Participants) | 28 | 34 | 27 | 24
  Day 28 | 18.0115 [7.1058 to 31.3329] | 20.3500 [7.3262 to 66.2388] | 18.9258 [7.6823 to 42.6557] | 17.4548 [9.0649 to 42.0806]

29. Primary Outcome: Apparent Total Clearance of SRT2104 From Plasma After Oral Administration (CL/F) on Day 1 and Day 28
Description: Blood samples were collected on Day 1 (pre-dose, 15 minutes, 30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 8 hour and 12 hour post-dose), Day 2 (24 hour post-Day 1 dose), Day 8 (pre-dose), Day 15 (pre-dose), Day 22 (pre-dose), Day 28 (pre-dose, and 15 minutes, 30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 8 hour and 12 hour post-dose) and Day 29 (24 hour post-Day 28 dose). The pre-dose sample was collected within one hour prior to study medication administration. The post-dose sample was collected within 2 minutes of the scheduled time. On Day 1 Day 2 and Day 29, participants fasted for at least 10 hour overnight.
Time Frame: as for outcome 26
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Liter/hour
Arm/Group | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 44 | 42 | 43
Liter/hour
  Day 1: number analyzed (Participants) | 28 | 36 | 30 | 27
  Day 1 | 494.0236 (625.5532) | 621.3930 (948.1533) | 1582.0131 (2707.3466) | 2181.8596 (2959.1044)
  Day 28: number analyzed (Participants) | 35 | 42 | 39 | 37
  Day 28 | 631.5519 (900.3648) | 956.6848 (2117.3623) | 1420.2734 (2128.7769) | 1887.2455 (2883.3080)

30. Primary Outcome: Apparent Volume of Distribution After Oral Administration (Vd/F) at Day 1 and Day 28
Description: as for outcome 29
Time Frame: as for outcome 26
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 44 | 42 | 43
mL/kg
  Day 1: number analyzed (Participants) | 28 | 36 | 30 | 27
  Day 1 | 12921.7880 (19802.8598) | 15767.2219 (29059.7570) | 38320.97415 (77339.06047) | 32262.5089 (45180.0346)
  Day 28: number analyzed (Participants) | 28 | 34 | 27 | 24
  Day 28 | 17509.8071 (27627.2504) | 48475.7739 (150725.4900) | 56531.7676 (108327.3925) | 51594.5474 (93165.0710)

31. Secondary Outcome: Mean Fasting Plasma Glucose (FPG) Levels Over Time
Description: The assessments were done at Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35 weekly at central laboratory. The analysis was reported for Day 8, Day 15, Day 22, Day 28 and Day 35.
Time Frame: Up to Day 35
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45
mmol per liter
  Day 8: number analyzed (Participants) | 43 | 42 | 42 | 41 | 40
  Day 8 | 10.46 (2.60) | 10.33 (2.30) | 11.10 (2.33) | 10.67 (2.19) | 10.37 (2.81)
  Day 15: number analyzed (Participants) | 41 | 37 | 43 | 40 | 40
  Day 15 | 10.08 (2.46) | 10.52 (2.40) | 10.51 (2.39) | 10.37 (2.30) | 10.41 (2.81)
  Day 22: number analyzed (Participants) | 42 | 37 | 43 | 38 | 40
  Day 22 | 10.03 (2.03) | 10.31 (2.66) | 11.24 (2.17) | 10.59 (2.35) | 10.56 (2.84)
  Day 28: number analyzed (Participants) | 43 | 36 | 42 | 38 | 38
  Day 28 | 9.60 (2.02) | 10.21 (2.12) | 10.49 (2.22) | 10.32 (2.16) | 10.05 (2.38)
  Day 35: number analyzed (Participants) | 41 | 41 | 43 | 39 | 42
  Day 35 | 10.10 (2.41) | 10.10 (2.21) | 9.92 (2.04) | 9.51 (2.62) | 9.03 (1.98)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day on Day 8 for FPG; Test type: Superiority; p = 0.997, ANOVA — Analysis was performed using ANOVA with Dunnett's test using the placebo group as the control, a 2-sided alpha of 0.05 was set as the significance threshold. No adjustments for covariates were made; Dunnett's test was used to control for inflation of alpha due to multiple comparisons, using the placebo group as the control
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day on Day 8 for FPG; Test type: Superiority; p = 0.581, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day on Day 8 for FPG; Test type: Superiority; p = 0.987, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day on Day 8 for FPG; Test type: Superiority; p = 0.999, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day on Day 15 for FPG; Test type: Superiority; p = 0.850, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day on Day 15 for FPG; Test type: Superiority; p = 0.843, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day on Day 15 for FPG; Test type: Superiority; p = 0.961, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day on Day 15 for FPG; Test type: Superiority; p = 0.939, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day on Day 22 for FPG; Test type: Superiority; p = 0.966, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day on Day 22 for FPG; Test type: Superiority; p = 0.075, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day on Day 22 for FPG; Test type: Superiority; p = 0.700, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day on Day 22 for FPG; Test type: Superiority; p = 0.732, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day on Day 28 for FPG; Test type: Superiority; p = 0.552, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 14: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day on Day 28 for FPG; Test type: Superiority; p = 0.196, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day on Day 28 for FPG; Test type: Superiority; p = 0.393, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day on Day 28 for FPG; Test type: Superiority; p = 0.775, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 17: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day on Day 35 for FPG; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 18: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day on Day 35 for FPG; Test type: Superiority; p = 0.989, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 19: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day on Day 35 for FPG; Test type: Superiority; p = 0.603, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 20: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day on Day 35 for FPG; Test type: Superiority; p = 0.108, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

32. Secondary Outcome: Change From Baseline in FPG Levels Over Time
Description: The assessments were done at Day 1, Day 8, Day 15, Day 22, Day 28 and Day 35 weekly at central laboratory. Baseline was defined as the assessment done on Day 1. The analysis was reported for Day 8, Day 15, Day 22, Day 28 and Day 35. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 8, Day 15, Day 22, Day 28 and Day 35) values.
Time Frame: Baseline (Day 1) and up to Day 35
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45
mmol per liter
  Day 8: number analyzed (Participants) | 43 | 41 | 41 | 39 | 40
  Day 8 | -0.30 (2.20) | -1.00 (3.23) | 0.16 (2.06) | -0.41 (2.77) | 0.17 (2.05)
  Day 15: number analyzed (Participants) | 41 | 36 | 42 | 38 | 40
  Day 15 | -0.72 (2.45) | -0.91 (2.61) | -0.41 (2.35) | -0.64 (2.78) | 0.17 (2.72)
  Day 22: number analyzed (Participants) | 42 | 37 | 42 | 37 | 40
  Day 22 | -0.74 (2.48) | -1.06 (3.63) | 0.28 (2.79) | -0.47 (2.90) | 0.40 (2.71)
  Day 28: number analyzed (Participants) | 43 | 35 | 42 | 36 | 38
  Day 28 | -1.17 (2.42) | -1.11 (3.45) | -0.52 (2.60) | -0.97 (2.83) | -0.15 (2.38)
  Day 35: number analyzed (Participants) | 41 | 39 | 43 | 37 | 42
  Day 35 | -0.73 (2.70) | -0.94 (2.47) | -1.24 (3.07) | -1.52 (3.29) | -1.14 (2.37)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in FPG on Day 8; Test type: Superiority; p = 0.525, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in FPG on Day 8; Test type: Superiority; p = 0.818, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in FPG on Day 8; Test type: Superiority; p = 0.999, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in FPG on Day 8; Test type: Superiority; p = 0.809, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in FPG on Day 15; Test type: Superiority; p = 0.993, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in FPG on Day 15; Test type: Superiority; p = 0.954, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in FPG on Day 15; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in FPG on Day 15; Test type: Superiority; p = 0.344, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in FPG on Day 22; Test type: Superiority; p = 0.968, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in FPG on Day 22; Test type: Superiority; p = 0.316, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in FPG on Day 22; Test type: Superiority; p = 0.984, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in FPG on Day 22; Test type: Superiority; p = 0.235, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in FPG on Day 28; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 14: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in FPG on Day 28; Test type: Superiority; p = 0.656, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in FPG on Day 28; Test type: Superiority; p = 0.994, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in FPG on Day 28; Test type: Superiority; p = 0.285, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 17: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in FPG on Day 35; Test type: Superiority; p = 0.992, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 18: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in FPG on Day 35; Test type: Superiority; p = 0.822, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 19: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in FPG on Day 35; Test type: Superiority; p = 0.538, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 20: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in FPG on Day 35; Test type: Superiority; p = 0.907, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

33. Secondary Outcome: Mean Fasting Plasma Insulin (FPI) Levels Over Time
Description: as for outcome 31
Time Frame: Up to Day 35
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45
mmol per liter
  Day 8: number analyzed (Participants) | 42 | 42 | 41 | 41 | 38
  Day 8 | 89.9 (59.63) | 92.3 (95.57) | 83.8 (52.19) | 74.5 (61.77) | 74.4 (51.36)
  Day 15: number analyzed (Participants) | 41 | 40 | 42 | 41 | 41
  Day 15 | 90.0 (70.89) | 78.4 (93.50) | 80.4 (45.86) | 80.5 (76.39) | 79.3 (89.05)
  Day 22: number analyzed (Participants) | 43 | 39 | 43 | 40 | 40
  Day 22 | 98.7 (98.55) | 74.3 (93.51) | 81.8 (47.79) | 78.8 (65.46) | 76.8 (57.34)
  Day 28: number analyzed (Participants) | 43 | 37 | 41 | 40 | 39
  Day 28 | 82.4 (56.91) | 91.7 (118.05) | 63.7 (44.87) | 63.3 (55.69) | 89.2 (134.56)
  Day 35: number analyzed (Participants) | 42 | 41 | 41 | 41 | 41
  Day 35 | 101.6 (70.49) | 110.5 (157.53) | 87.1 (56.22) | 84.0 (78.95) | 115.3 (213.37)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day on Day 8 for FPI; Test type: Superiority; p = 0.999, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day on Day 8 for FPI; Test type: Superiority; p = 0.982, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day on Day 8 for FPI; Test type: Superiority; p = 0.677, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day on Day 8 for FPI; Test type: Superiority; p = 0.688, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day on Day 15 for FPI; Test type: Superiority; p = 0.903, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day on Day 15 for FPI; Test type: Superiority; p = 0.945, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day on Day 15 for FPI; Test type: Superiority; p = 0.949, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day on Day 15 for FPI; Test type: Superiority; p = 0.924, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day on Day 22 for FPI; Test type: Superiority; p = 0.394, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day on Day 22 for FPI; Test type: Superiority; p = 0.687, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day on Day 22 for FPI; Test type: Superiority; p = 0.568, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day on Day 22 for FPI; Test type: Superiority; p = 0.486, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day on Day 28 for FPI; Test type: Superiority; p = 0.973, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 14: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day on Day 28 for FPI; Test type: Superiority; p = 0.739, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day on Day 28 for FPI; Test type: Superiority; p = 0.731, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day on Day 28 for FPI; Test type: Superiority; p = 0.991, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 17: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day on Day 35 for FPI; Test type: Superiority; p = 0.994, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 18: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day on Day 35 for FPI; Test type: Superiority; p = 0.963, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 19: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day on Day 35 for FPI; Test type: Superiority; p = 0.929, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 20: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day on Day 35 for FPI; Test type: Superiority; p = 0.970, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

34. Secondary Outcome: Change From Baseline in FPI Over Time
Description: as for outcome 32
Time Frame: Baseline (Day 1) and up to Day 35
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45
mmol per liter
  Day 8: number analyzed (Participants) | 40 | 42 | 37 | 39 | 36
  Day 8 | 7.2 (66.75) | 12.2 (80.20) | 12.3 (49.91) | 12.9 (63.97) | 4.7 (37.72)
  Day 15: number analyzed (Participants) | 39 | 39 | 39 | 39 | 8
  Day 15 | 10.8 (77.13) | -6.5 (48.51) | 8.1 (45.43) | 18.8 (88.06) | 8.3 (96.60)
  Day 22: number analyzed (Participants) | 41 | 38 | 40 | 38 | 37
  Day 22 | 17.6 (90.89) | -4.6 (55.62) | 10.6 (56.34) | 20.2 (75.69) | 0.3 (49.95)
  Day 28: number analyzed (Participants) | 41 | 36 | 39 | 38 | 36
  Day 28 | 1.0 (51.66) | 8.9 (95.04) | -6.9 (41.45) | 4.1 (57.16) | 15.2 (138.79)
  Day 35: number analyzed (Participants) | 40 | 40 | 40 | 39 | 38
  Day 35 | 20.4 (80.92) | 30.7 (103.55) | 13.7 (47.92) | 22.3 (79.42) | 48.0 (216.64)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in FPI on Day 8; Test type: Superiority; p = 0.989, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in FPI on Day 8; Test type: Superiority; p = 0.989, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in FPI on Day 8; Test type: Superiority; p = 0.982, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in FPI on Day 8; Test type: Superiority; p = 0.999, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in FPI on Day 15; Test type: Superiority; p = 0.685, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in FPI on Day 15; Test type: Superiority; p = 0.999, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in FPI on Day 15; Test type: Superiority; p = 0.971, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in FPI on Day 15; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in FPI on Day 22; Test type: Superiority; p = 0.405, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in FPI on Day 22; Test type: Superiority; p = 0.975, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in FPI on Day 22; Test type: Superiority; p = 0.999, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in FPI on Day 22; Test type: Superiority; p = 0.629, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in FPI on Day 28; Test type: Superiority; p = 0.982, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 14: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in FPI on Day 28; Test type: Superiority; p = 0.982, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in FPI on Day 28; Test type: Superiority; p = 0.999, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in FPI on Day 28; Test type: Superiority; p = 0.874, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 17: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in FPI on Day 35; Test type: Superiority; p = 0.986, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 18: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in FPI on Day 35; Test type: Superiority; p = 0.997, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 19: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in FPI on Day 35; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 20: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in FPI on Day 35; Test type: Superiority; p = 0.697, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

35. Secondary Outcome: Mean Post-prandial Glucose (PPG) and Post-prandial Insulin (PPI) Levels at Day 28
Description: The assessment of PPG and PPI was performed on Day 28 at 30 minutes, 60 minutes and 2 hour after the participant consumed the standardized meal (morning breakfast).
Time Frame: Day 28
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45
mmol per liter
  PPG, 30 minutes: number analyzed (Participants) | 24 | 26 | 28 | 27 | 26
  PPG, 30 minutes | 12.91 (2.94) | 12.95 (2.66) | 13.58 (3.05) | 13.12 (2.90) | 11.41 (2.77)
  PPG, 60 minutes: number analyzed (Participants) | 24 | 26 | 29 | 27 | 26
  PPG, 60 minutes | 14.05 (3.13) | 14.05 (3.57) | 15.44 (3.05) | 14.77 (3.16) | 13.08 (3.70)
  PPG, 2 hour: number analyzed (Participants) | 43 | 35 | 41 | 40 | 39
  PPG, 2 hour | 13.16 (4.26) | 13.15 (3.55) | 14.74 (3.15) | 13.90 (3.60) | 13.61 (4.43)
  PPI, 30 minutes: number analyzed (Participants) | 24 | 26 | 28 | 28 | 26
  PPI, 30 minutes | 237.6 (222.95) | 217.2 (198.91) | 188.3 (172.53) | 160.2 (153.46) | 163.0 (179.83)
  PPI, 60 minutes: number analyzed (Participants) | 24 | 26 | 28 | 27 | 26
  PPI, 60 minutes | 298.1 (232.43) | 285.4 (339.90) | 223.0 (167.72) | 189.2 (145.83) | 226.6 (200.82)
  PPI, 2 hour: number analyzed (Participants) | 43 | 37 | 40 | 40 | 39
  PPI, 2 hour | 224.4 (129.69) | 215.0 (309.78) | 192.5 (132.93) | 183.8 (160.20) | 206.4 (202.40)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day at 30 minutes for PPG; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day at 30 minutes for PPG; Test type: Superiority; p = 0.812, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day at 30 minutes for PPG; Test type: Superiority; p = 0.996, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day at 30 minutes for PPG; Test type: Superiority; p = 0.198, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day at 60 minutes for PPG; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day at 60 minutes for PPG; Test type: Superiority; p = 0.358, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day at 60 minutes for PPG; Test type: Superiority; p = 0.852, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day at 60 minutes for PPG; Test type: Superiority; p = 0.678, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day at 2 hour for PPG; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day at 2 hour for PPG; Test type: Superiority; p = 0.191, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day at 2 hour for PPG; Test type: Superiority; p = 0.805, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day at 2 hour for PPG; Test type: Superiority; p = 0.960, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day at 30 minutes for PPI; Test type: Superiority; p = 0.985, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 14: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day at 30 minutes for PPI; Test type: Superiority; p = 0.733, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day at 30 minutes for PPI; Test type: Superiority; p = 0.365, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day at 30 minutes for PPI; Test type: Superiority; p = 0.413, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 17: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day at 60 minutes for PPI; Test type: Superiority; p = 0.765, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 18: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day at 60 minutes for PPI; Test type: Superiority; p = 0.434, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 19: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day at 60 minutes for PPI; Test type: Superiority; p = 0.184, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 20: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day at 60 minutes for PPI; Test type: Superiority; p = 0.142, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 21: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day at 2 hour for PPI; Test type: Superiority; p = 0.999, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 22: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day at 2 hour for PPI; Test type: Superiority; p = 0.876, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 23: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day at 2 hour for PPI; Test type: Superiority; p = 0.756, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 24: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day at 2 hour for PPI; Test type: Superiority; p = 0.983, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

36. Secondary Outcome: Change From Baseline in PPG and PPI Levels at Day 28
Description: The assessment of PPG and PPI was performed at 30 minutes, 60 minutes and 2 hour after the participant consumed the standardized meal (morning breakfast) on Day 1 and Day 28. Baseline for PPG was defined as the assessment value of FPG done on Day 1 and Baseline for PPI was defined as the assessment value of FPI done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (30 min, 60 min and 2 h at Day 28) values.
Time Frame: Baseline (Day 1) and Day 28
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45
mmol per liter
  PPG, 30 minutes: number analyzed (Participants) | 24 | 26 | 28 | 25 | 26
  PPG, 30 minutes | 3.38 (2.85) | 2.82 (2.40) | 3.40 (2.52) | 3.14 (1.75) | 2.00 (2.17)
  PPG, 60 minutes: number analyzed (Participants) | 24 | 26 | 29 | 25 | 26
  PPG, 60 minutes | 4.53 (2.86) | 3.92 (3.55) | 5.12 (2.57) | 4.74 (2.34) | 3.68 (3.08)
  PPG, 2 hour: number analyzed (Participants) | 43 | 35 | 41 | 38 | 38
  PPG, 2 hour | 3.56 (3.37) | 2.93 (3.33) | 4.23 (2.88) | 3.66 (2.54) | 3.47 (3.44)
  PPI, 30 minutes: number analyzed (Participants) | 24 | 26 | 28 | 28 | 26
  PPI, 30 minutes | 162.4 (204.29) | 108.7 (136.13) | 119.2 (157.32) | 94.9 (109.96) | 57.4 (73.07)
  PPI, 60 minutes: number analyzed (Participants) | 24 | 26 | 28 | 27 | 26
  PPI, 60 minutes | 222.9 (206.99) | 176.9 (278.91) | 153.9 (146.74) | 128.4 (105.95) | 121.0 (95.22)
  PPI, 2 hour: number analyzed (Participants) | 43 | 37 | 40 | 40 | 39
  PPI, 2 hour | 142.0 (113.58) | 123.3 (253.84) | 128.7 (106.87) | 120.5 (129.95) | 117.3 (127.26)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in PPG at 30 minutes; Test type: Superiority; p = 0.809, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in PPG at 30 minutes; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in PPG at 30 minutes; Test type: Superiority; p = 0.989, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in PPG at 30 minutes; Test type: Superiority; p = 0.130, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in PPG at 60 minutes; Test type: Superiority; p = 0.870, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in PPG at 60 minutes; Test type: Superiority; p = 0.864, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in PPG at 60 minutes; Test type: Superiority; p = 0.997, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in PPG at 60 minutes; Test type: Superiority; p = 0.682, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in PPG at 2 hour; Test type: Superiority; p = 0.798, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in PPG at 2 hour; Test type: Superiority; p = 0.730, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in PPG at 2 hour; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in PPG at 2 hour; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in PPI at 30 minutes; Test type: Superiority; p = 0.464, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 14: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in PPI at 30 minutes; Test type: Superiority; p = 0.634, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in PPI at 30 minutes; Test type: Superiority; p = 0.254, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in PPI at 30 minutes; Test type: Superiority; p = 0.034, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 17: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in PPI at 60 minutes; Test type: Superiority; p = 0.765, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 18: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in PPI at 60 minutes; Test type: Superiority; p = 0.434, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 19: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in PPI at 60 minutes; Test type: Superiority; p = 0.184, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 20: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in PPI at 60 minutes; Test type: Superiority; p = 0.142, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 21: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day for change from Baseline in PPI at 2 hour; Test type: Superiority; p = 0.955, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 22: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day for change from Baseline in PPI at 2 hour; Test type: Superiority; p = 0.985, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 23: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day for change from Baseline in PPI at 2 hour; Test type: Superiority; p = 0.923, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 24: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day for change from Baseline in PPI at 2 hour; Test type: Superiority; p = 0.883, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

37. Secondary Outcome: Mean Glycosylated Hemoglobin A (HbA1c) Levels on Day 28
Description: The sample for HbA1c assessment was collected on Day 28. HbA1c is used to show how well their diabetes is being controlled in participants with diabetes. The HbA1c test gives the average blood glucose levels over the pervious two to three months.
Time Frame: Day 28
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 36 | 42 | 40 | 40
Percentage of HbA1c | 8.18 (0.95) | 8.66 (1.00) | 8.64 (0.93) | 8.54 (1.16) | 8.29 (0.90)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Test type: Superiority; p = 0.118, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Test type: Superiority; p = 0.119, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Test type: Superiority; p = 0.293, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Test type: Superiority; p = 0.966, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

38. Secondary Outcome: Change From Baseline in HbA1c Levels at Day 28
Description: HbA1c is used to show how well their diabetes is being controlled in participants with diabetes. The HbA1c test gives the average blood glucose levels over the pervious two to three months. The sample for HbA1c assessment was collected on Day 1 and Day 28. Baseline value was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 28) value.
Time Frame: Baseline (Day 1) and Day 28
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 43 | 35 | 42 | 38 | 40
Percentage of HbA1c | -0.31 (0.55) | -0.23 (0.68) | -0.05 (0.52) | 0.01 (0.78) | -0.10 (0.71)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Test type: Superiority; p = 0.940, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Test type: Superiority; p = 0.197, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Test type: Superiority; p = 0.097, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Test type: Superiority; p = 0.404, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

39. Secondary Outcome: AUC From Time 0 to 1 h (AUC 0-1) and AUC From Time 0 to 2 h (AUC 0-2) for PPG and PPI at Day 1 and Day 28
Description: The assessment of PPG and PPI was performed at 30 minutes, 60 minnutes and 2 hour after the participant consumed the standardized meal (morning breakfast) on Day 1 and Day 28. AUC with respect to these time interval was calculated using the linear trapezoidal rule by the sum of the areas between each chronological pair of assessments (using observed times) for PPG and PPI.
Time Frame: Day 1 (30 minutes, 60 minutes and 2 hour) and Day 28 (30 minutes, 60 minutes and 2 hour)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol*hour per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 30 | 31 | 32 | 31 | 30
mmol*hour per liter
  Day 1, AUC 0-1, PPG: number analyzed (Participants) | 25 | 26 | 29 | 25 | 26
  Day 1, AUC 0-1, PPG | 13.10 (2.69) | 14.08 (3.40) | 14.28 (3.50) | 14.43 (4.18) | 12.68 (2.73)
  Day 28, AUC 0-1, PPG: number analyzed (Participants) | 24 | 26 | 28 | 25 | 26
  Day 28, AUC 0-1, PPG | 12.35 (2.45) | 12.52 (2.41) | 13.25 (2.58) | 12.92 (2.27) | 11.33 (2.63)
  Day 1, AUC 0-2, PPG: number analyzed (Participants) | 27 | 27 | 28 | 27 | 27
  Day 1, AUC 0-2, PPG | 27.39 (5.72) | 29.35 (7.64) | 29.87 (7.20) | 29.95 (9.34) | 26.07 (5.99)
  Day 28, AUC 0-2, PPG: number analyzed (Participants) | 28 | 25 | 28 | 27 | 26
  Day 28, AUC 0-2, PPG | 25.89 (5.84) | 25.98 (5.64) | 28.30 (5.51) | 27.01 (5.11) | 24.14 (6.40)
  Day 1, AUC 0-1, PPI: number analyzed (Participants) | 24 | 28 | 28 | 26 | 24
  Day 1, AUC 0-1, PPI | 192.4 (121.08) | 211.1 (245.53) | 176.6 (105.51) | 168.3 (123.33) | 186.0 (92.55)
  Day 28, AUC 0-1, PPI: number analyzed (Participants) | 24 | 26 | 27 | 27 | 26
  Day 28, AUC 0-1, PPI | 212.1 (176.25) | 207.1 (202.43) | 168.1 (135.71) | 138.8 (120.34) | 164.6 (175.64)
  Day 1, AUC 0-2, PPI: number analyzed (Participants) | 26 | 28 | 26 | 28 | 25
  Day 1, AUC 0-2, PPI | 423.8 (289.68) | 478.8 (584.46) | 418.4 (251.25) | 377.6 (297.27) | 385.8 (167.81)
  Day 28, AUC 0-2, PPI: number analyzed (Participants) | 28 | 26 | 27 | 29 | 26
  Day 28, AUC 0-2, PPI | 444.8 (332.82) | 477.7 (538.49) | 394.5 (276.65) | 334.7 (256.51) | 381.3 (378.70)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day of AUC 0-1 at Day 1 for PPG; Test type: Superiority; p = 0.2060, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day of AUC 0-1 at Day 1 for PPG; Test type: Superiority; p = 0.1790, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day of AUC 0-1 at Day 1 for PPG; Test type: Superiority; p = 0.2741, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day of AUC 0-1 at Day 1 for PPG; Test type: Superiority; p = 0.6001, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 5: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day of AUC 0-1 at Day 28 for PPG; Test type: Superiority; p = 0.6711, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 6: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day of AUC 0-1 at Day 28 for PPG; Test type: Other; p = 0.1361, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 7: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day of AUC 0-1 at Day 28 for PPG; Test type: Superiority; p = 0.3369, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 8: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day of AUC 0-1 at Day 28 for PPG; Test type: Superiority; p = 0.0975, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 9: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day of AUC 0-2 at Day 1 for PPG; Test type: Superiority; p = 0.2184, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 10: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day of AUC 0-2 at Day 1 for PPG; Test type: Superiority; p = 0.1013, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 11: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day of AUC 0-2 at Day 1 for PPG; Test type: Superiority; p = 0.3286, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 12: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day of AUC 0-2 at Day 1 for PPG; Test type: Superiority; p = 0.5193, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 13: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day of AUC 0-2 at Day 28 for PPG; Test type: Superiority; p = 0.9788, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 14: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day of AUC 0-2 at Day 28 for PPG; Test type: Superiority; p = 0.1214, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 15: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day of AUC 0-2 at Day 28 for PPG; Test type: Superiority; p = 0.5751, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 16: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day of AUC 0-2 at Day 28 for PPG; Test type: Superiority; p = 0.2409, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 17: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day of AUC 0-1 at Day 1 for PPI; Test type: Superiority; p = 0.4829, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 18: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day of AUC 0-1 at Day 1 for PPI; Test type: Superiority; p = 0.7563, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 19: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day of AUC 0-1 at Day 1 for PPI; Test type: Superiority; p = 0.2907, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 20: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day of AUC 0-1 at Day 1 for PPI; Test type: Superiority; p = 0.7663, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 21: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day of AUC 0-1 at Day 28 for PPI; Test type: Superiority; p = 0.5825, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 22: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day of AUC 0-1 at Day 28 for PPI; Test type: Superiority; p = 0.3220, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 23: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day of AUC 0-1 at Day 28 for PPI; Test type: Superiority; p = 0.0564, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 24: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 0.25 g/day of AUC 0-1 at Day 28 for PPI; Test type: Superiority; p = 0.1960, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 25: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day of AUC 0-2 at Day 1 for PPI; Test type: Superiority; p = 0.5997, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 26: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day of AUC 0-2 at Day 1 for PPI; Test type: Superiority; p = 0.9637, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 27: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day of AUC 0-2 at Day 1 for PPI; Test type: Superiority; p = 0.3240, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 28: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day of AUC 0-2 at Day 1 for PPI; Test type: Superiority; p = 0.8440, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 29: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day of AUC 0-2 at Day 28 for PPI; Test type: Superiority; p = 0.6483, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 30: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day of AUC 0-2 at Day 28 for PPI; Test type: Superiority; p = 0.6452, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 31: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day of AUC 0-2 at Day 28 for PPI; Test type: Superiority; p = 0.1253, Wilcoxon test — No adjustments for covariates were made
Statistical Analysis 32: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day of AUC 0-2 at Day 28 for PPI; Test type: Superiority; p = 0.2583, Wilcoxon test — No adjustments for covariates were made

40. Secondary Outcome: Mean Fructosamine Levels at Day 1 and Day 28
Description: Fructosamine (a glycated protein) level enables assessment of long-term glycemic control in participants with diabetes mellitus. The blood samples for fructosamine assessment was obtained at Day 1 and Day 28.
Time Frame: Day 1 and Day 28
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45
mmol/L
  Day 1 | 320.07 (61.28) | 320.38 (49.20) | 319.82 (56.73) | 328.44 (62.90) | 296.00 (41.86)
  Day 28 | 305.70 (56.04) | 315.97 (60.46) | 330.15 (61.32) | 318.63 (50.90) | 285.28 (57.45)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day at Day 1 for fructosamine; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day at Day 1 for fructosamine; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day at Day 1 for fructosamine; Test type: Superiority; p = 0.901, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day at Day 1 for fructosamine; Test type: Superiority; p = 0.155, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day at Day 28 for fructosamine; Test type: Superiority; p = 0.845, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day at Day 28 for fructosamine; Test type: Superiority; p = 0.164, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day at Day 28 for fructosamine; Test type: Superiority; p = 0.699, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day at Day 28 for fructosamine; Test type: Superiority; p = 0.313, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

41. Secondary Outcome: Change From Baseline in Fructosamine Levels at Day 28
Description: Fructosamine (a glycated protein) level enables assessment of long-term glycemic control in participants with diabetes mellitus. The blood samples for fructosamine assessment was obtained at Day 1 and Day 28. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 28) value.
Time Frame: Baseline (Day 1) and Day 28
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: mmol per liter
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45
mmol per liter | -14.37 (41.18) | -6.67 (40.27) | 9.76 (62.77) | -4.68 (44.64) | -2.14 (48.83)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Test type: Superiority; p = 0.896, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Test type: Superiority; p = 0.080, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Test type: Superiority; p = 0.792, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Test type: Superiority; p = 0.645, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

42. Secondary Outcome: Mean Homeostatic Model Assessment-insulin Resistance (HOMA-IR) at Day 1 and Day 28
Description: HOMA-IR was derived from FPG and FPI as: FPI (micro units [mU]/mL)*FPG (mmol per liter) divided by 22.5. HOMA-IR was calculated from the Day 1 and Day 28 FPG and FPI values at Day 1 and Day 28.
Time Frame: Day 1 and Day 28
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mU*mmol per liter^2
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45
mU*mmol per liter^2
  Day 1: number analyzed (Participants) | 41 | 40 | 41 | 39 | 40
  Day 1 | 5.4 (3.98) | 5.7 (5.45) | 5.2 (5.20) | 4.1 (3.31) | 5.0 (3.75)
  Day 28: number analyzed (Participants) | 43 | 36 | 41 | 38 | 38
  Day 28 | 4.9 (3.56) | 5.9 (7.28) | 3.9 (2.55) | 4.0 (3.66) | 5.9 (10.10)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day at Day 1 for HOMA-IR; Test type: Superiority; p = 0.992, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day at Day 1 for HOMA-IR; Test type: Superiority; p = 0.999, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day at Day 1 for HOMA-IR; Test type: Superiority; p = 0.548, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day at Day 1 for HOMA-IR; Test type: Superiority; p = 0.989, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day at Day 28 for HOMA-IR; Test type: Superiority; p = 0.877, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day at Day 28 for HOMA-IR; Test type: Superiority; p = 0.887, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day at Day 28 for HOMA-IR; Test type: Superiority; p = 0.916, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day at Day 28 for HOMA-IR; Test type: Superiority; p = 0.860, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

43. Secondary Outcome: Change From Baseline in HOMA-IR at Day 28
Description: HOMA-IR was derived from FPG and FPI as: FPI (mU/mL)*FPG (mmol per liter) divided by 22.5. HOMA-IR was calculated from the Day 1 and Day 28 FPG and FPI values at Day 1 and Day 28. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 28) value.
Time Frame: Baseline (Day 1) and Day 28
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mU*mmol per liter^2
Groups:
- Placebo: Participants received oral dose of matching placebo to SRT2104 capsule, once daily for 28 consecutive days. The study medication was administered as 8 capsules per day to maintain the blinding, at the same time every morning, approximately 15-30 minutes following the start of meal consumption with 1 to 2 glasses of water.
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 41 | 34 | 39 | 35 | 35
mU*mmol per liter^2 | -0.4 (3.61) | 0.0 (7.26) | -0.9 (3.47) | -0.1 (3.83) | 1.0 (10.17)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Test type: Superiority; p = 0.996, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Test type: Superiority; p = 0.989, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Test type: Superiority; p = 0.999, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Test type: Superiority; p = 0.763, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

44. Secondary Outcome: Mean HOMA-percentage Cell Beta Function at Day 1 and Day 28
Description: HOMA-percentage cell beta function was derived from FPG and FPI as: 20*FPI (mU/mL) divided by FPG (mmol per liter) minus 3.5. HOMA-percentage cell beta function was calculated from the Day 1 and Day 28 FPG and FPI values at Day 1 and Day 28.
Time Frame: Day 1 and Day 28
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of beta cell function
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 46 | 45 | 46 | 45 | 45
Percentage of beta cell function
  Day 1: number analyzed (Participants) | 41 | 40 | 41 | 39 | 40
  Day 1 | 38.3 (38.15) | 31.8 (46.38) | 31.2 (35.46) | 27.2 (21.39) | 30.2 (23.03)
  Day 28: number analyzed (Participants) | 43 | 36 | 41 | 38 | 38
  Day 28 | 42.9 (34.71) | 42.9 (57.90) | 32.6 (34.57) | 28.4 (26.48) | 40.9 (48.31)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day at Day 1 for HOMA-percentage of beta cell function; Test type: Superiority; p = 0.810, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day at Day 1 for HOMA-percentage of beta cell function; Test type: Superiority; p = 0.753, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day at Day 1 for HOMA-percentage of beta cell function; Test type: Superiority; p = 0.404, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day at Day 1 for HOMA-percentage of beta cell function; Test type: Superiority; p = 0.671, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs SRT2104 0.25 g/Day; Placebo versus SRT2104 0.25 g/day at Day 28 for HOMA-percentage of beta cell function; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs SRT2104 0.5 g/Day; Placebo versus SRT2104 0.5 g/day at Day 28 for HOMA-percentage of beta cell function; Test type: Superiority; p = 0.622, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs SRT2104 1.0 g/Day; Placebo versus SRT2104 1.0 g/day at Day 28 for HOMA-percentage of beta cell function; Test type: Superiority; p = 0.332, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs SRT2104 2.0 g/Day; Placebo versus SRT2104 2.0 g/day at Day 28 for HOMA-percentage of beta cell function; Test type: Superiority; p = 0.998, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

45. Secondary Outcome: Change From Baseline in HOMA-percentage of Beta Cell Function at Day 28
Description: HOMA-percentage cell beta function was derived from FPG and FPI as: 20*FPI (mU/mL) divided by FPG (mmol per liter) minus 3.5. HOMA-percentage cell beta function was calculated from the Day 1 and Day 28 FPG and FPI values at Day 1 and Day 28. Baseline was defined as assessment done on Day 1. Baseline was defined as the assessment done on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1) from the individual post-Baseline (Day 28) value.
Time Frame: Baseline (Day 1) and Day 28
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of beta cell function
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
Number analyzed (Participants) | 41 | 34 | 39 | 35 | 35
Percentage of beta cell function | 5.8 (34.02) | 8.5 (42.09) | 2.3 (17.87) | 3.1 (26.45) | 7.6 (51.96)
Statistical Analysis 1: Comparison: Placebo vs SRT2104 0.25 g/Day; Test type: Superiority; p = 0.994, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs SRT2104 0.5 g/Day; Test type: Superiority; p = 0.979, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SRT2104 1.0 g/Day; Test type: Superiority; p = 0.993, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs SRT2104 2.0 g/Day; Test type: Superiority; p = 0.999, ANOVA — [p-value comment as in outcome 31, analysis 1]; [statistical method as in outcome 31, analysis 1]

ADVERSE EVENTS:
Time Frame: AE's and SAE's were collected from the start of study medication (Day 1) up to Follow-up (58 days)
Description: Safety Analysis Set Population was used.
Arm/Group | Placebo | SRT2104 0.25 g/Day | SRT2104 0.5 g/Day | SRT2104 1.0 g/Day | SRT2104 2.0 g/Day
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 1/44 | 0/42 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 1/43 | 1/44 | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 7/43 | 4/43 | 12/44 | 5/42 | 8/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | SRT2104 0.25 g/Day (N=43) | SRT2104 0.5 g/Day (N=44) | SRT2104 1.0 g/Day (N=42) | SRT2104 2.0 g/Day (N=43)
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | SRT2104 0.25 g/Day (N=43) | SRT2104 0.5 g/Day (N=44) | SRT2104 1.0 g/Day (N=42) | SRT2104 2.0 g/Day (N=43)
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 4 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 3 | 4 | 1 | 2
Asthenia (General disorders) | 1 | 1 | 4 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 3 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.